CLINICAL TRIAL: NCT02969525
Title: A Multicenter, Phase 2B, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Evaluate the Efficacy and Safety of Bimekizumab in Active Psoriatic Arthritis
Brief Title: A Study to Evaluate the Dose Response Based on the Efficacy, Safety and Tolerability of Bimekizumab in Subjects With Active Psoriatic Arthritis Which is a Type of Inflammatory Arthritis
Acronym: BE ACTIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA0008; 2016-001103-23 (EudraCT Number)
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; PsA; Bimekizumab
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Subjects will receive for 12 Weeks Placebo and will then be re-randomized to Bimekizumab dosage regimen 2 or Bimekizumab dosage regimen 3 for 36 Weeks.
  Interventions: Other: Placebo
- Bimekizumab dosage regimen 1 (Experimental): Subjects will receive for 12 Weeks Bimekizumab dosage regimen 1 and will then be re-randomized to Bimekizumab dosage regimen 2 or Bimekizumab dosage regimen 3 for 36 Weeks.
  Interventions: Drug: Bimekizumab
- Bimekizumab dosage regimen 2 (Experimental): Subjects will receive for 48 Weeks Bimekizumab dosage regimen 2.
  Interventions: Drug: Bimekizumab
- Bimekizumab dosage regimen 3 (Experimental): Subjects will receive for 48 Weeks Bimekizumab dosage regimen 3.
  Interventions: Drug: Bimekizumab
- Bimekizumab dosage regimen 4 (Experimental): Subjects will receive for 12 Weeks Bimekizumab dosage regimen 4 and will then be re-randomized to Bimekizumab dosage regimen 2 for 36 Weeks.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Other: Placebo
  Arms: Placebo
Drug: Bimekizumab — Bimekizumab in different dosage regimens.
  Other Names: UCB4940
  Arms: Bimekizumab dosage regimen 1; Bimekizumab dosage regimen 2; Bimekizumab dosage regimen 3; Bimekizumab dosage regimen 4

SUMMARY:
This is a study to evaluate the dose response based on the efficacy, safety and tolerability of bimekizumab in subjects with active psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a documented diagnosis of adult-onset PsA classified by Classification Criteria for Psoriatic Arthritis (CASPAR) criteria with symptoms for at least 6 months prior to Screening, with active psoriatic arthritis (PsA) at Baseline/Day 1, and must have at Baseline tender joint count (TJC) >=3 out of 78 and swollen joint count (SJC) >=3 out of 76
* Subject must be rheumatoid factor and anti-cyclic citrullinated peptide (CCP) antibodies negative
* Subject must have active psoriatic lesion(s) and/or a documented history of psoriasis
* Subjects who are regularly taking nonsteroidal anti-inflammatory drug (NSAIDs)/COX-2 inhibitors as part of their PsA therapy are required to be on a stable dose/dose regimen for at least 14 days before Baseline
* Subjects taking corticosteroids must be on an average daily dose of <=10mg/day prednisone or equivalent for at least 14 days before Baseline and should remain on a stable dose through the Week 16 visit
* Subjects taking methotrexate (MTX) (<=25mg /week) are allowed to continue their medication if started at least 12 weeks prior to Baseline, with a stable dose for at least 8 weeks before randomization
* Subjects taking leflunomide (LEF; <=20mg/day or an average of 20mg/day if not dosed daily) are allowed to continue their medication if started at least 3 months prior to Baseline, with a stable dose for at least 8 weeks before randomization. Dose and dosing schedule should remain stable up to Week 16
* Subjects may be tumor necrosis factor (TNF) inhibitor naïve or may have received 1 prior TNF inhibitor. Subjects who have been on a TNF inhibitor previously must have:

  1. experienced an inadequate response to previous treatment given for at least 3 months
  2. been intolerant to administration (eg, had a side-effect/adverse event (AE) that led to discontinuation)
  3. lost access to TNF inhibitor for other reasons

Exclusion Criteria:

* Subjects with any current sign or symptom that may indicate an active infection (with the exception of the common cold) or has had an infection requiring systemic antibiotics within 2 weeks of Baseline/Day 1
* Subjects with a history of chronic or recurrent infections, or a serious or life-threatening infection within the 6 months prior to the Baseline Visit
* Subjects with concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Subjects with known history of or current clinically active infection with Histoplasma, Coccidioides, Paracoccidioides, Pneumocystis, Blastomyces, or Aspergillus or current active Candidiasis
* Subjects receiving any live (includes attenuated) vaccination within the 8 weeks prior to Baseline
* Subjects with known tuberculosis (TB) infection, at high risk of acquiring TB infection, with latent TB infection (LTBI), or current or history of nontuberculous mycobacteria (NTMB) infection
* Subjects with a diagnosis of inflammatory conditions other than psoriasis or psoriatic arthritis
* Subjects with concurrent malignancy or a history of malignancy during the past 5 years will be excluded, with following exceptions that may be included:

  1. <= 3 excised or ablated basal cell carcinomas of the skin
  2. One squamous cell carcinoma of the skin (stage T1 maximum) successfully excised, or ablated only (other treatments, ie, chemotherapy, do not apply), with no signs of recurrence or metastases for more than 2 years prior to Screening
  3. Actinic keratosis (-es)
  4. Squamous cell carcinoma-in-situ of the skin successfully excised, or ablated, more than 6 months prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273(UCB)
Locations (40):
- United States (13):
  - Pa0008 007, San Diego, California
  - Pa0008 005, Aventura, Florida
  - Pa0008 003, Hagerstown, Maryland
  - Pa0008 011, Lansing, Minnesota
  - Pa0008 025, Lexington, New York
  - Pa0008 014, Portland, Oregon
  - Pa0008 001, Duncansville, Pennsylvania
  - Pa0008 012, Johnston, Rhode Island
  - Pa0008 004, Charleston, South Carolina
  - Pa0008 010, Jackson, Tennessee
  - Pa0008 006, Dallas, Texas
  - Pa0008 013, Mesquite, Texas
  - Pa0008 002, Seattle, Washington
- Czechia (7):
  - Pa0008 205, Brno
  - Pa0008 207, Olomouc
  - Pa0008 201, Prague
  - Pa0008 202, Prague
  - Pa0008 209, Prague
  - Pa0008 210, Prague
  - Pa0008 203, Zlín
- Germany (4):
  - Pa0008 302, Cologne
  - Pa0008 309, Erlangen
  - Pa0008 304, Hamburg
  - Pa0008 301, Ratingen
- Hungary (2):
  - Pa0008 403, Budakeszierdő
  - Pa0008 401, Veszprém
- Poland (9):
  - Pa0008 452, Bialystok
  - Pa0008 453, Elblag
  - Pa0008 456, Elblag
  - Pa0008 455, Krakow
  - Pa0008 451, Poznan
  - Pa0008 450, Torun
  - Pa0008 454, Warsaw
  - Pa0008 459, Warsaw
  - Pa0008 465, Wroclaw
- Russia (5):
  - Pa0008 604, Moscow
  - Pa0008 605, Moscow
  - Pa0008 607, Moscow
  - Pa0008 606, Saint Petersburg
  - Pa0008 608, Saint Petersburg

REFERENCES:
- [Result] Mease PJ, Asahina A, Gladman DD, Tanaka Y, Tillett W, Ink B, Assudani D, de la Loge C, Coarse J, Eells J, Gossec L. Effect of bimekizumab on symptoms and impact of disease in patients with psoriatic arthritis over 3 years: results from BE ACTIVE. Rheumatology (Oxford). 2023 Feb 1;62(2):617-628. doi: 10.1093/rheumatology/keac353. PMID 35789257
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794
- [Derived] Ritchlin CT, Kavanaugh A, Merola JF, Schett G, Scher JU, Warren RB, Gottlieb AB, Assudani D, Bedford-Rice K, Coarse J, Ink B, McInnes IB. Bimekizumab in patients with active psoriatic arthritis: results from a 48-week, randomised, double-blind, placebo-controlled, dose-ranging phase 2b trial. Lancet. 2020 Feb 8;395(10222):427-440. doi: 10.1016/S0140-6736(19)33161-7. PMID 32035552

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in October 2016 and concluded in July 2018.
Pre-assignment Details: The study included a 28-Day Screening Period, followed by a Double-blind Period from Day 1 to Week 12, prior to treatment re-randomization, a Dose-blind Period, from Week 12 after the treatment re-randomization and up to Week 48 and a Safety Follow-Up (SFU) Period, post week 48.
  The Participant Flow refers to the Randomized Set and Dose-Blind Set.
Groups:
- Placebo: Participants received Placebo during the 12 Weeks Double-Blind Period.
- BKZ 16 mg: Participants received Bimekizumab (BKZ) 16 milligrams (mg) every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period.
- BKZ 160 mg: Participants received Bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period followed by the same dose during the 36 Weeks Dose-Blind Period.
- BKZ 160 mg LD: Participants received Bimekizumab (BKZ) 320 mg at Baseline followed by 160 mg every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period.
- BKZ 320 mg: Participants received Bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period followed by the same dose during the 36 Weeks Dose-Blind Period.
- Placebo - BKZ 160 mg: After the 12 Weeks Double-Blind Period participants randomized to Placebo were re-randomized to receive Bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) for 36 weeks in the Dose-Blind Period.
- Placebo - BZK 320 mg: After the 12 Weeks Double-Blind Period participants randomized to Placebo were re-randomized to receive Bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) for 36 weeks in the Dose-Blind Period.
- BKZ 16 mg - BKZ 160 mg: After the 12 Weeks Double-Blind Period participants randomized to Bimekizumab (BKZ) 16 mg every 4 weeks (Q4W) were re-randomized to receive BKZ 160 mg Q4W for 36 weeks in the Dose-Blind Period.
- BZK 16 mg - BZK 320 mg: After the 12 Weeks Double-Blind Period participants randomized to Bimekizumab (BKZ) 16 mg every 4 weeks (Q4W) were re-randomized to receive BKZ 320 mg Q4W for 36 weeks in the Dose-Blind Period.
- BZK 160 mg LD - BZK 160 mg: After the 12 Weeks Double-Blind Period participants randomized to Bimekizumab (BKZ) 320 mg at Baseline followed by 160 mg every 4 weeks (Q4W) were re-randomized to receive BKZ 160 mg Q4W for 36 weeks in the Dose-Blind Period.
- BZK 160 mg - BKZ Dose 160 mg: After the 12 Weeks Double-Blind Period participants randomized to Bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) were re-randomized to receive BKZ 160 mg Q4W for 36 weeks in the Dose-Blind Period.
- BKZ 320 mg - BKZ 320 mg: After the 12 Weeks Double-Blind Period participants randomized to Bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) were re-randomized to receive BKZ 320 mg Q4W for 36 weeks in the Dose-Blind Period.
Period: Double-Blind Period
Arm/Group | Placebo | BKZ 16 mg | BKZ 160 mg | BKZ 160 mg LD | BKZ 320 mg | Placebo - BKZ 160 mg | Placebo - BZK 320 mg | BKZ 16 mg - BKZ 160 mg | BZK 16 mg - BZK 320 mg | BZK 160 mg LD - BZK 160 mg | BZK 160 mg - BKZ Dose 160 mg | BKZ 320 mg - BKZ 320 mg
Started | 42 | 41 | 41 | 41 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Double-Blind Period | 42 | 41 | 40 | 39 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Wk12 and Started Dose-Blind | 40 | 41 | 40 | 37 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 40 | 41 | 40 | 37 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — LOW EGFR | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study medication discontinued prior Wk12 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose-Blind Period
Arm/Group | Placebo | BKZ 16 mg | BKZ 160 mg | BKZ 160 mg LD | BKZ 320 mg | Placebo - BKZ 160 mg | Placebo - BZK 320 mg | BKZ 16 mg - BKZ 160 mg | BZK 16 mg - BZK 320 mg | BZK 160 mg LD - BZK 160 mg | BZK 160 mg - BKZ Dose 160 mg | BKZ 320 mg - BKZ 320 mg
Started | 0 | 0 | 0 | 0 | 0 | 20 | 20 | 22 | 19 | 37 | 40 | 41
Completed | 0 | 0 | 0 | 0 | 0 | 20 | 18 | 22 | 18 | 34 | 38 | 39
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0
Not completed — Non-cooperating patient | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrew before Safety Follow-up visit | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refer to the Full Analysis Set (FAS), which consisted of all randomized study participants who received at least 1 dose of investigational medicinal product (IMP) and had a valid measurement of the primary efficacy variable at Baseline.
Arm/Group | Placebo | BKZ 16 mg | BKZ 160 mg | BKZ 160 mg LD | BKZ 320 mg | Total Title
Number analyzed (Participants) | 42 | 41 | 41 | 41 | 41 | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 35 | 40 | 36 | 36 | 185
  >=65 years | 4 | 6 | 1 | 5 | 5 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.02 (12.07) | 49.98 (13.56) | 48.00 (11.65) | 49.05 (12.99) | 50.39 (12.08) | 49.29 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 21 | 27 | 18 | 101
  Male | 24 | 24 | 20 | 14 | 23 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Black | 1 | 1 | 2 | 1 | 0 | 5
  White | 40 | 40 | 39 | 40 | 41 | 200

OUTCOME MEASURES:

1. Primary Outcome: ACR50 (American College of Rheumatology 50% Improvement) Response at Week 12
Description: The ACR50 response rate was based on 50% improvement relative to Baseline in the following measures:
  * Tender Joint Count (TJC) based on 78 joints
  * Swollen Joint Count (SJC) based on 76 joints
  * 3 of the 5 remaining core set measures:
    * Disease activity as assessed by Patient's Global Assessment of Disease Activity (PGADA)
    * Disease activity as assessed by Physician's Global Assessment of Disease Activity (PhGADA)
    * Pain as assessed by Patient's Assessment of Arthritis Pain (PtAAP)
    * Physical function as assessed by Health Assessment Questionnaire - Disability Index (HAQ-DI)
    * Acute phase response as assessed by high sensitivity C-reactive protein (hs CRP).
Time Frame: Week 12
Population: The Full Analysis Set (FAS) consisted of all randomized study participants who received at least 1 dose of investigational medicinal product (IMP) and had a valid measurement of the primary efficacy variable at Baseline.
Measure: Number; unit: percentage of subjects
Groups:
- Placebo (FAS): Participants received Placebo during the 12 Weeks Double-Blind Period, forming the Full Analysis Set (FAS).
- BKZ 16 mg (FAS): Participants received Bimekizumab (BKZ) 16 milligrams (mg) every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period, forming the Full Analysis Set (FAS).
- BKZ 160 mg (FAS): Participants received Bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period followed by the same dose during the 36 Weeks Dose-Blind Period, forming the Full Analysis Set (FAS).
- BKZ 160 mg LD (FAS): Participants received Bimekizumab (BKZ) 320 mg at Baseline followed by 160 mg every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period, forming the Full Analysis Set (FAS).
- BKZ 320 mg (FAS): Participants received Bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period followed by the same dose during the 36 Weeks Dose-Blind Period, forming the Full Analysis Set (FAS).
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 160 mg (FAS) | BKZ 160 mg LD (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 42 | 41 | 41 | 41 | 41
percentage of subjects | 7.1 | 26.8 | 41.5 | 46.3 | 24.4
Statistical Analysis 1: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS) vs BKZ 160 mg (FAS) vs BKZ 160 mg LD (FAS) vs BKZ 320 mg (FAS); Statistic and p-value were calculated using a Cochran-Mantel-Haenszel test (test for non-zero correlation statistic) based on modified ridit scores and including geographic region and prior Tumor Necrosis Factor (TNF) inhibitor exposure as stratification factors. The 160 loading dose arm was not considered in the dose-response because this is a mixed dose and the test is examining linear dose response; Test type: Other; p = 0.031, Cochran-Mantel-Haenszel; Correlation statistic = 4.6
Statistical Analysis 2: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS); For differences in relation to placebo: Odds Ratio, confidence interval, and p-value were derived from a logistic regression model including fixed effects for treatment, geographic region and prior Tumor Factor Necrosis (TNF) inhibitor exposure; Test type: Other — The pairwise testing of each bimekizumab dose versus placebo accounted for multiplicity by using a fixed sequence testing procedure with each bimekizumab dose being tested sequentially from the highest dose to the lowest dose. If the sequential testing failed to reach significance at a significance level of alpha=0.05, then the pairwise testing continued and the comparison was seen as non-significant; p = 0.032, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 4.2, 95% CI 2-sided [1.13 to 15.23]
Statistical Analysis 3: Comparison: Placebo (FAS) vs BKZ 160 mg (FAS); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 8.1, 95% CI 2-sided [2.28 to 28.74]
Statistical Analysis 4: Comparison: Placebo (FAS) vs BKZ 160 mg LD (FAS); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; p < 0.001, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 9.7, 95% CI 2-sided [2.73 to 34.26]
Statistical Analysis 5: Comparison: Placebo (FAS) vs BKZ 320 mg (FAS); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.051, Regression, Logistic — The p-values were displayed as nominal p-values; Odds Ratio (OR) = 3.7, 95% CI 2-sided [1.00 to 13.68]

2. Secondary Outcome: ACR20 (American College of Rheumatology 20% Improvement) Response at Week 12
Description: The ACR20 response rate was based on 20% improvement relative to Baseline in the following measures:
  * TJC based on 78 joints
  * SJC based on 76 joints
  * 3 of the 5 remaining core set measures:
    * Disease activity as assessed by PGADA
    * Disease activity as assessed by PhGADA
    * Pain as assessed by PtAAP
    * Physical function as assessed by HAQ-DI
    * Acute phase response as assessed by hs CRP
  Note: Nonresponder imputation was used to account for missing data in the primary analysis, the study participants with a missing ACR score at Week 12 or who discontinued IMP prior to the Week 12 Visit were considered nonresponders for the primary analysis.
Time Frame: Week 12
Population: The FAS consisted of all randomized study participants who received at least 1 dose of IMP and had a valid measurement of the primary efficacy variable at Baseline.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 160 mg (FAS) | BKZ 160 mg LD (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 42 | 41 | 41 | 41 | 41
percentage of subjects | 19.0 | 53.7 | 73.2 | 61.0 | 51.2
Statistical Analysis 1: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS); For differences in relation to Placebo: Odds Ratio, confidence interval, and p-value were derived from a logistic regression model including fixed effects for treatment, geographic region and prior Tumor Necrosis Factor (TNF) inhibitor exposure; Test type: Other; p = 0.002, Regression, Logistic — No sequential testing procedure was used for the secondary efficacy variables. The p-values were displayed as nominal p-values; Odds Ratio (OR) = 4.6, 95% CI 2-sided [1.73 to 12.39]
Statistical Analysis 2: Comparison: Placebo (FAS) vs BKZ 160 mg (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 11.0, 95% CI 2-sided [3.91 to 30.95]
Statistical Analysis 3: Comparison: Placebo (FAS) vs BKZ 160 mg LD (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 6.2, 95% CI 2-sided [2.31 to 16.84]
Statistical Analysis 4: Comparison: Placebo (FAS) vs BKZ 320 mg (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.004, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 4.2, 95% CI 2-sided [1.59 to 11.35]

3. Secondary Outcome: ACR70 (American College of Rheumatology 70% Improvement) Response at Week 12
Description: The ACR70 response rate was based on 70% improvement relative to Baseline in the following measures:
  * TJC based on 78 joints
  * SJC based on 76 joints
  * 3 of the 5 remaining core set measures:
    * Disease activity as assessed by PGADA
    * Disease activity as assessed by PhGADA
    * Pain as assessed by PtAAP
    * Physical function as assessed by HAQ-DI
    * Acute phase response as assessed by hs CRP
  Note: Nonresponder imputation was used to account for missing data in the primary analysis, the study participants with a missing ACR score at Week 12 or who discontinued IMP prior to the Week 12 Visit were considered nonresponders for the primary analysis.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 160 mg (FAS) | BKZ 160 mg LD (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 42 | 41 | 41 | 41 | 41
percentage of subjects | 4.8 | 12.2 | 19.5 | 31.7 | 14.6
Statistical Analysis 1: Comparison: Placebo (FAS) vs BKZ 16 mg (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.279, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.4, 95% CI 2-sided [0.50 to 11.31]
Statistical Analysis 2: Comparison: Placebo (FAS) vs BKZ 160 mg (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.065, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 4.1, 95% CI 2-sided [0.92 to 17.88]
Statistical Analysis 3: Comparison: Placebo (FAS) vs BKZ 160 mg LD (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.006, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 7.5, 95% CI 2-sided [1.77 to 31.28]
Statistical Analysis 4: Comparison: Placebo (FAS) vs BKZ 320 mg (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.172, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.9, 95% CI 2-sided [0.63 to 13.39]

4. Secondary Outcome: PASI90 (Psoriasis Area Severity Index) Response at Week 12 in the Subgroup of Subjects With Psoriasis Involving at Least 3 % Body Surface Area (BSA) at Baseline/Day 1
Description: The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked).
  Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 12
Population: Subset of of study participants in the FAS with at least (≥) 3 percent (%) psoriasis (PSO) Body Surface Area (BSA) at Baseline (NRI).
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 160 mg (FAS) | BKZ 160 mg LD (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 20 | 14 | 16 | 17 | 11
percentage of subjects | 10.0 | 35.7 | 62.5 | 52.9 | 45.5

5. Secondary Outcome: PASI75 (Psoriasis Area Severity Index) Response at Week 12 in the Subgroup of Subjects With Psoriasis Involving at Least 3 % Body Surface Area (BSA) at Baseline/Day 1
Description: The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked).
  Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (FAS) | BKZ 16 mg (FAS) | BKZ 160 mg (FAS) | BKZ 160 mg LD (FAS) | BKZ 320 mg (FAS)
Number analyzed (Participants) | 20 | 14 | 16 | 17 | 11
percentage of subjects | 10.0 | 57.1 | 68.8 | 70.6 | 72.7

6. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During the Study
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP.
Time Frame: From Screening Period until the Safety Follow-Up Visit (up to Week 72)
Population: The Safety Set (SS) consisted of all randomized study participants who received at least 1 dose of IMP. The 160mg LD group and 160mg groups are combined into one column to see the effect of the 160mg dose overall.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (SS) - up to Wk 12: This arm consisted of all participants who received Placebo at any time in the study (up to Week 12). Participants formed the Safety Set (SS).
- BKZ 16 mg (SS) - up to Wk 12: This arm consisted of all participants who received Bimekizumab (BKZ) 16 milligrams (mg) every 4 weeks (Q4W) at any time in the study (up to Week 12). Participants formed the SS.
- BKZ 160 mg & 160 mg LD (SS) - up to Wk 68: This arm consisted of all participants who received Bimekizumab (BKZ) 320 mg at Baseline followed by 160 mg every 4 weeks (Q4W) and Bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) at any time in the study (up to Week 68). Participants formed the SS.
- BKZ 320 mg (SS) - up to Wk 68: This arm consisted of all participants who received Bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) at any time in the study (up to Week 68). Participants formed the SS.
Arm/Group | Placebo (SS) - up to Wk 12 | BKZ 16 mg (SS) - up to Wk 12 | BKZ 160 mg & 160 mg LD (SS) - up to Wk 68 | BKZ 320 mg (SS) - up to Wk 68
Number analyzed (Participants) | 42 | 39 | 126 | 80
percentage of participants | 57.1 | 33.33 | 74.6 | 72.5

7. Secondary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE) During the Study
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Screening Period until the Safety Follow-Up Visit (up to Week 72)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) - up to Wk 12 | BKZ 16 mg (SS) - up to Wk 12 | BKZ 160 mg & 160 mg LD (SS) - up to Wk 68 | BKZ 320 mg (SS) - up to Wk 68
Number analyzed (Participants) | 42 | 39 | 126 | 80
percentage of participants | 2.4 | 0 | 6.3 | 0

8. Secondary Outcome: Percentage of Participants Who Withdrew Due to an Adverse Event (AE) During the Study
Description: as for outcome 6
Time Frame: From Screening Period until the Safety Follow-Up Visit (up to Week 72)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) - up to Wk 12 | BKZ 16 mg (SS) - up to Wk 12 | BKZ 160 mg & 160 mg LD (SS) - up to Wk 68 | BKZ 320 mg (SS) - up to Wk 68
Number analyzed (Participants) | 42 | 39 | 126 | 80
percentage of participants | 4.8 | 0 | 4.8 | 2.5

9. Secondary Outcome: Changes From Baseline in Vital Signs During the Study (Diastolic Blood Pressure, Systolic Blood Pressure)
Description: Diastolic and systolic blood pressure were measured in millimeters of mercury (mmHg).
Time Frame: Baseline, 30 min and 1 hour post dose, Week 1, Week 2, pre- and post dose for the following Weeks: 4, 8, 12, 16, 20, 24, 28, 32, 36, 40 and 44 and Week 48
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo (SS): Participants received Placebo during the 12 Weeks Double-Blind Period, forming the Safety Set (SS).
- BKZ 16 mg (SS): Participants received Bimekizumab (BKZ) 16 milligrams (mg) every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period, forming the SS.
- BKZ 160 mg (SS): Participants received Bimekizumab (BKZ) 160 mg every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period followed by the same dose during the 36 Weeks Dose-Blind Period, forming the SS.
- BKZ 160 mg LD (SS): Participants received Bimekizumab (BKZ) 320 mg at Baseline followed by 160 mg every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period, forming the SS.
- BKZ 320 mg (SS): Participants received Bimekizumab (BKZ) 320 mg every 4 weeks (Q4W) during the 12 Weeks Double-Blind Period followed by the same dose during the 36 Weeks Dose-Blind Period, forming the SS.
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
mmHg
  Diastolic Blood Pressure 30 min post dose | 1.3 (8.9) | -1.2 (4.9) | -1.2 (5.4) | 0.6 (6.1) | -0.6 (5.3)
  Diastolic Blood Pressure 1 h post dose | 1.1 (8.8) | -2.0 (6.3) | -0.7 (8.1) | 1.2 (6.7) | -1.0 (5.5)
  Diastolic Blood Pressure Week 1: number analyzed (Participants) | 41 | 39 | 43 | 41 | 41
  Diastolic Blood Pressure Week 1 | 0.1 (9.6) | -0.3 (6.5) | 0.6 (11.4) | -0.9 (6.6) | -0.4 (6.5)
  Diastolic Blood Pressure Week 2 | 0.7 (10.4) | -0.7 (6.5) | -1.0 (8.9) | -2.7 (8.3) | -0.1 (9.0)
  Diastolic Blood Pressure Week 4 pre-dose: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Diastolic Blood Pressure Week 4 pre-dose | 0.0 (8.2) | -1.7 (8.4) | -1.4 (10.7) | -0.8 (7.8) | -1.3 (7.4)
  Diastolic Blood Pressure Week 4 post dose: number analyzed (Participants) | 41 | 39 | 41 | 40 | 40
  Diastolic Blood Pressure Week 4 post dose | -2.0 (8.7) | -1.0 (7.3) | -1.2 (8.9) | -0.9 (8.3) | -1.6 (7.6)
  Diastolic Blood Pressure Week 8 pre-dose: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Diastolic Blood Pressure Week 8 pre-dose | 1.0 (8.2) | -1.3 (8.7) | 0.3 (8.7) | -0.5 (7.0) | 0.2 (6.9)
  Diastolic Blood Pressure Week 8 post dose: number analyzed (Participants) | 41 | 39 | 42 | 39 | 41
  Diastolic Blood Pressure Week 8 post dose | -0.9 (9.1) | -1.1 (8.4) | 0.6 (8.7) | -0.7 (7.3) | -2.2 (7.4)
  Diastolic Blood Pressure Week 12 pre-dose: number analyzed (Participants) | 42 | 39 | 42 | 39 | 41
  Diastolic Blood Pressure Week 12 pre-dose | 0.2 (9.1) | -1.1 (10.4) | 0.2 (8.5) | -1.5 (7.9) | -0.6 (8.2)
  Diastolic Blood Pressure Week 12 post dose: number analyzed (Participants) | 40 | 39 | 42 | 37 | 41
  Diastolic Blood Pressure Week 12 post dose | -0.3 (9.6) | -2.0 (10.0) | 0.3 (8.3) | -1.8 (7.9) | -2.6 (8.0)
  Diastolic Blood Pressure Week 16 pre-dose: number analyzed (Participants) | 42 | 39 | 42 | 38 | 41
  Diastolic Blood Pressure Week 16 pre-dose | -2.7 (9.6) | -3.5 (8.9) | -0.8 (8.6) | -1.2 (8.7) | -0.4 (7.9)
  Diastolic Blood Pressure Week 16 post dose: number analyzed (Participants) | 40 | 39 | 39 | 36 | 39
  Diastolic Blood Pressure Week 16 post dose | -3.0 (9.1) | -1.9 (8.3) | -1.7 (9.2) | -1.1 (7.9) | -2.4 (8.7)
  Diastolic Blood Pressure Week 20 pre-dose: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Diastolic Blood Pressure Week 20 pre-dose | 0.5 (10.3) | -1.8 (9.0) | -0.6 (8.3) | -1.4 (8.3) | -1.8 (7.3)
  Diastolic Blood Pressure Week 20 post dose: number analyzed (Participants) | 39 | 39 | 38 | 36 | 40
  Diastolic Blood Pressure Week 20 post dose | 0.1 (9.5) | -3.1 (8.3) | -0.4 (9.2) | -3.0 (9.3) | -2.6 (7.1)
  Diastolic Blood Pressure Week 24 pre-dose: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Diastolic Blood Pressure Week 24 pre-dose | -0.4 (7.6) | -1.6 (7.2) | -0.7 (9.3) | 1.0 (6.9) | -1.0 (6.6)
  Diastolic Blood Pressure Week 24 post dose: number analyzed (Participants) | 39 | 38 | 38 | 35 | 39
  Diastolic Blood Pressure Week 24 post dose | -0.6 (7.5) | -1.7 (7.9) | -0.3 (8.2) | -0.3 (7.6) | -1.4 (7.9)
  Diastolic Blood Pressure Week 28 pre-dose: number analyzed (Participants) | 39 | 39 | 41 | 35 | 40
  Diastolic Blood Pressure Week 28 pre-dose | 1.4 (7.9) | -0.6 (9.7) | 0.9 (9.5) | -0.6 (6.9) | -0.5 (7.5)
  Diastolic Blood Pressure Week 28 post dose: number analyzed (Participants) | 38 | 39 | 39 | 34 | 39
  Diastolic Blood Pressure Week 28 post dose | 1.2 (8.7) | -2.0 (9.4) | 1.2 (9.0) | -0.2 (7.1) | -1.8 (7.1)
  Diastolic Blood Pressure Week 32 pre-dose: number analyzed (Participants) | 39 | 39 | 40 | 35 | 39
  Diastolic Blood Pressure Week 32 pre-dose | 0.2 (8.5) | -1.7 (8.6) | 1.6 (9.2) | -0.3 (9.3) | -1.2 (8.6)
  Diastolic Blood Pressure Week 32 post dose: number analyzed (Participants) | 36 | 39 | 37 | 34 | 39
  Diastolic Blood Pressure Week 32 post dose | 0.7 (10.0) | -3.0 (8.6) | 0.1 (9.6) | -0.6 (8.5) | -2.1 (8.5)
  Diastolic Blood Pressure Week 36 pre-dose: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Diastolic Blood Pressure Week 36 pre-dose | 0.0 (8.6) | -0.6 (9.2) | 1.4 (8.9) | -0.9 (7.2) | 0.8 (7.5)
  Diastolic Blood Pressure Week 36 post dose: number analyzed (Participants) | 37 | 38 | 38 | 31 | 38
  Diastolic Blood Pressure Week 36 post dose | 1.6 (7.7) | -1.6 (9.2) | 1.3 (9.3) | -1.7 (6.8) | -0.1 (7.1)
  Diastolic Blood Pressure Week 40 pre-dose: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Diastolic Blood Pressure Week 40 pre-dose | 0.8 (7.6) | -2.5 (9.7) | 1.0 (9.5) | -1.0 (7.2) | -1.9 (6.8)
  Diastolic Blood Pressure Week 40 post dose: number analyzed (Participants) | 37 | 38 | 40 | 33 | 37
  Diastolic Blood Pressure Week 40 post dose | 0.9 (7.7) | -1.8 (9.1) | 0.2 (8.3) | -0.8 (6.6) | -0.1 (7.3)
  Diastolic Blood Pressure Week 44 pre-dose: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Diastolic Blood Pressure Week 44 pre-dose | 1.4 (9.3) | -2.1 (7.7) | 1.3 (9.2) | -0.4 (6.7) | -2.4 (10.9)
  Diastolic Blood Pressure Week 44 post dose: number analyzed (Participants) | 36 | 38 | 40 | 33 | 39
  Diastolic Blood Pressure Week 44 post dose | 2.3 (9.2) | -1.3 (7.6) | -0.7 (8.7) | -1.4 (8.1) | -1.5 (6.5)
  Diastolic Blood Pressure Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Diastolic Blood Pressure Week 48 | 1.8 (9.2) | 0.4 (9.7) | 1.1 (9.1) | 0.6 (8.7) | -0.8 (6.4)
  Systolic Blood Pressure 30 min post dose | 0.8 (8.1) | 0.5 (9.7) | -0.8 (8.2) | 1.5 (8.8) | -2.5 (9.7)
  Systolic Blood Pressure 1 hour post dose | -0.6 (9.4) | -2.0 (10.5) | 0.2 (8.7) | 1.0 (8.4) | -1.8 (7.1)
  Systolic Blood Pressure Week 1: number analyzed (Participants) | 41 | 39 | 43 | 41 | 41
  Systolic Blood Pressure Week 1 | -1.7 (10.8) | -1.3 (10.0) | 1.7 (12.9) | -2.4 (8.3) | -1.6 (11.0)
  Systolic Blood Pressure Week 2 | -0.7 (12.9) | -0.2 (9.8) | -0.1 (13.2) | -2.7 (8.2) | -0.4 (11.9)
  Systolic Blood Pressure Week 4 pre-dose: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Systolic Blood Pressure Week 4 pre-dose | -2.6 (11.4) | -1.5 (10.6) | -1.0 (13.0) | -2.3 (10.5) | -2.7 (11.2)
  Systolic Blood Pressure Week 4 post dose: number analyzed (Participants) | 41 | 39 | 41 | 40 | 40
  Systolic Blood Pressure Week 4 post dose | -3.5 (12.1) | -0.6 (10.4) | -2.2 (11.8) | -0.6 (9.1) | -3.7 (11.3)
  Systolic Blood Pressure Week 8 pre-dose: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Systolic Blood Pressure Week 8 pre-dose | -2.1 (13.1) | -0.8 (10.7) | -1.1 (11.3) | -3.6 (11.7) | -1.3 (10.4)
  Systolic Blood Pressure Week 8 post dose: number analyzed (Participants) | 41 | 39 | 42 | 39 | 41
  Systolic Blood Pressure Week 8 post dose | -3.2 (12.6) | -1.9 (11.6) | -0.3 (11.1) | -2.8 (10.2) | -1.9 (12.0)
  Systolic Blood Pressure Week 12 pre-dose: number analyzed (Participants) | 42 | 39 | 42 | 39 | 41
  Systolic Blood Pressure Week 12 pre-dose | -3.3 (12.4) | 1.6 (13.7) | -3.1 (11.7) | -4.4 (10.8) | -2.6 (9.7)
  Systolic Blood Pressure Week 12 post dose: number analyzed (Participants) | 40 | 39 | 42 | 37 | 41
  Systolic Blood Pressure Week 12 post dose | -3.9 (14.1) | 2.1 (11.1) | -1.9 (12.0) | -3.6 (10.1) | -2.4 (10.1)
  Systolic Blood Pressure Week 16 pre-dose: number analyzed (Participants) | 42 | 39 | 42 | 38 | 41
  Systolic Blood Pressure Week 16 pre-dose | -3.6 (15.1) | -2.3 (12.3) | -4.3 (11.3) | -4.3 (12.5) | -2.3 (11.4)
  Systolic Blood Pressure Week 16 post dose: number analyzed (Participants) | 40 | 39 | 39 | 36 | 39
  Systolic Blood Pressure Week 16 post dose | -3.7 (17.1) | -2.6 (11.7) | -3.4 (12.7) | -2.7 (11.0) | -5.7 (8.5)
  Systolic Blood Pressure Week 20 pre-dose: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Systolic Blood Pressure Week 20 pre-dose | -2.0 (13.1) | -3.2 (12.5) | -2.6 (11.9) | -5.4 (9.7) | -4.5 (10.5)
  Systolic Blood Pressure Week 20 post dose: number analyzed (Participants) | 39 | 39 | 38 | 36 | 40
  Systolic Blood Pressure Week 20 post dose | -1.9 (14.5) | -3.2 (13.0) | -3.7 (12.2) | -7.9 (11.9) | -4.4 (9.9)
  Systolic Blood Pressure Week 24 pre-dose: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Systolic Blood Pressure Week 24 pre-dose | -3.1 (10.5) | -1.1 (9.5) | -2.7 (12.3) | -3.6 (10.1) | -0.3 (10.5)
  Systolic Blood Pressure Week 24 post dose: number analyzed (Participants) | 39 | 38 | 38 | 35 | 39
  Systolic Blood Pressure Week 24 post dose | -2.6 (10.9) | -2.8 (10.5) | -2.2 (11.7) | -3.0 (9.7) | -1.1 (10.5)
  Systolic Blood Pressure Week 28 pre-dose: number analyzed (Participants) | 39 | 39 | 41 | 35 | 40
  Systolic Blood Pressure Week 28 pre-dose | -0.1 (11.4) | -2.5 (12.8) | -2.5 (13.1) | 0.4 (11.6) | -2.9 (11.3)
  Systolic Blood Pressure Week 28 post dose: number analyzed (Participants) | 38 | 39 | 39 | 34 | 39
  Systolic Blood Pressure Week 28 post dose | -1.1 (12.1) | -2.9 (11.1) | -2.6 (12.4) | -0.7 (11.9) | -4.6 (11.2)
  Systolic Blood Pressure Week 32 pre-dose: number analyzed (Participants) | 39 | 39 | 40 | 35 | 39
  Systolic Blood Pressure Week 32 pre-dose | -0.9 (13.1) | -1.5 (13.3) | -0.6 (12.4) | 0.6 (11.0) | -3.7 (12.4)
  Systolic Blood Pressure Week 32 post dose: number analyzed (Participants) | 36 | 39 | 37 | 34 | 39
  Systolic Blood Pressure Week 32 post dose | -1.7 (12.6) | -2.2 (11.6) | 0.3 (12.5) | -0.4 (11.1) | -4.8 (10.6)
  Systolic Blood Pressure Week 36 pre-dose: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Systolic Blood Pressure Week 36 pre-dose | -3.1 (11.9) | 1.1 (13.9) | -0.2 (13.6) | -1.8 (11.2) | -3.2 (11.1)
  Systolic Blood Pressure Week 36 post dose: number analyzed (Participants) | 37 | 38 | 38 | 31 | 38
  Systolic Blood Pressure Week 36 post dose | -0.6 (11.1) | 1.3 (12.6) | -0.5 (12.4) | -3.8 (10.8) | -3.8 (11.4)
  Systolic Blood Pressure Week 40 pre-dose: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Systolic Blood Pressure Week 40 pre-dose | -3.3 (12.1) | -3.1 (11.4) | -1.6 (12.9) | -4.0 (9.5) | -1.2 (11.0)
  Systolic Blood Pressure Week 40 post dose: number analyzed (Participants) | 37 | 38 | 40 | 33 | 37
  Systolic Blood Pressure Week 40 post dose | -2.3 (11.7) | -0.4 (12.7) | -1.2 (13.8) | -3.2 (11.6) | -2.2 (9.6)
  Systolic Blood Pressure Week 44 pre-dose: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Systolic Blood Pressure Week 44 pre-dose | -2.8 (12.3) | -2.8 (9.9) | 0.0 (13.1) | -5.1 (9.9) | -3.9 (10.3)
  Systolic Blood Pressure Week 44 post dose: number analyzed (Participants) | 36 | 38 | 40 | 33 | 39
  Systolic Blood Pressure Week 44 post dose | -1.8 (14.5) | -1.2 (9.5) | -0.6 (10.4) | -4.6 (10.3) | -3.8 (10.5)
  Systolic Blood Pressure Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Systolic Blood Pressure Week 48 | -1.1 (14.0) | -0.1 (12.5) | -0.1 (12.6) | -2.8 (11.5) | -5.2 (9.6)

10. Secondary Outcome: Changes From Baseline in Vital Signs During the Study (Pulse Rate)
Description: Pulse rate was measured in beats per minute (beats/min).
Time Frame: as for outcome 9
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
beats/min
  30 min post dose | 0.4 (5.4) | -0.8 (5.6) | -1.5 (7.2) | -2.3 (7.5) | -1.1 (7.2)
  1 hour post dose | 0.3 (6.7) | 1.0 (11.3) | -0.8 (7.6) | -0.8 (8.1) | -0.4 (7.0)
  Week 1: number analyzed (Participants) | 41 | 39 | 43 | 41 | 41
  Week 1 | 2.9 (8.3) | -1.5 (7.5) | -0.7 (7.1) | 0.6 (8.9) | -0.8 (9.0)
  Week 2 | 1.2 (6.4) | -1.7 (5.7) | -0.7 (7.9) | -1.0 (9.1) | -0.4 (6.9)
  Week 4 pre-dose: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Week 4 pre-dose | -0.2 (5.3) | -2.1 (6.9) | -1.9 (8.1) | 0.1 (9.8) | -1.0 (6.6)
  Week 4 post dose: number analyzed (Participants) | 41 | 39 | 41 | 40 | 40
  Week 4 post dose | 0.4 (8.6) | -2.6 (6.6) | -2.7 (9.5) | -0.5 (9.4) | -1.1 (6.2)
  Week 8 pre-dose: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Week 8 pre-dose | 0.9 (6.5) | -0.6 (8.0) | -1.6 (8.6) | 0.8 (6.9) | -1.3 (8.2)
  Week 8 post dose: number analyzed (Participants) | 41 | 39 | 42 | 39 | 41
  Week 8 post dose | -0.1 (6.9) | -1.3 (8.6) | -1.9 (8.6) | 0.0 (8.5) | -2.3 (8.3)
  Week 12 pre-dose: number analyzed (Participants) | 42 | 39 | 42 | 39 | 41
  Week 12 pre-dose | 1.1 (10.2) | -2.2 (8.5) | -2.9 (10.5) | -1.7 (9.5) | -1.1 (8.4)
  Week 12 post dose: number analyzed (Participants) | 40 | 39 | 42 | 37 | 41
  Week 12 post dose | -0.6 (8.8) | -3.3 (8.8) | -3.6 (9.4) | -2.1 (9.7) | -2.0 (7.8)
  Week 16 pre-dose: number analyzed (Participants) | 42 | 39 | 42 | 38 | 41
  Week 16 pre-dose | -0.2 (8.5) | -2.1 (5.8) | -2.9 (8.0) | -1.9 (10.1) | -1.3 (7.2)
  Week 16 post dose: number analyzed (Participants) | 40 | 39 | 39 | 36 | 39
  Week 16 post dose | -0.1 (9.9) | -3.5 (5.5) | -3.7 (9.7) | -2.1 (9.8) | -2.2 (7.3)
  Week 20 pre-dose: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Week 20 pre-dose | -0.1 (10.3) | -2.4 (7.0) | -1.7 (10.3) | 0.0 (9.0) | -1.2 (9.0)
  Week 20 post dose: number analyzed (Participants) | 39 | 39 | 38 | 36 | 40
  Week 20 post dose | -0.7 (6.8) | -2.3 (7.8) | -2.1 (9.7) | -0.1 (8.5) | -1.3 (8.9)
  Week 24 pre-dose: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Week 24 pre-dose | -0.5 (7.9) | -2.0 (8.1) | -2.8 (10.4) | -0.7 (7.3) | -1.2 (7.8)
  Week 24 post dose: number analyzed (Participants) | 39 | 38 | 38 | 35 | 39
  Week 24 post dose | -0.9 (7.8) | -2.9 (8.5) | -3.0 (9.6) | -1.3 (6.9) | -2.5 (7.1)
  Week 28 pre-dose: number analyzed (Participants) | 39 | 39 | 41 | 35 | 40
  Week 28 pre-dose | 1.9 (9.7) | -2.1 (10.0) | 0.0 (9.3) | -0.5 (11.2) | 0.2 (8.3)
  Week 28 post dose: number analyzed (Participants) | 38 | 39 | 39 | 34 | 39
  Week 28 post dose | 1.8 (7.5) | -3.0 (9.4) | -0.5 (8.5) | -0.8 (10.0) | 0.0 (7.5)
  Week 32 pre-dose: number analyzed (Participants) | 39 | 39 | 40 | 35 | 39
  Week 32 pre-dose | 3.3 (10.0) | -0.9 (7.9) | -2.0 (9.2) | -1.2 (10.6) | -0.3 (7.8)
  Week 32 post dose: number analyzed (Participants) | 36 | 39 | 37 | 34 | 39
  Week 32 post dose | 3.3 (8.4) | -0.8 (7.8) | -3.0 (9.5) | -1.9 (9.6) | -2.0 (8.8)
  Week 36 pre-dose: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Week 36 pre-dose | 0.7 (8.5) | 0.2 (7.5) | -2.6 (8.6) | -2.6 (10.2) | -0.5 (9.7)
  Week 36 post dose: number analyzed (Participants) | 37 | 38 | 38 | 31 | 38
  Week 36 post dose | 1.1 (7.6) | -0.8 (8.2) | -3.0 (9.8) | -2.5 (8.2) | -1.4 (9.6)
  Week 40 pre-dose: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Week 40 pre-dose | 2.7 (10.3) | -0.5 (8.8) | 1.0 (10.1) | -1.7 (7.6) | 2.0 (9.4)
  Week 40 post dose: number analyzed (Participants) | 37 | 38 | 40 | 33 | 37
  Week 40 post dose | 0.9 (8.3) | -1.7 (8.3) | 0.0 (8.9) | -2.0 (8.4) | 0.5 (9.1)
  Week 44 pre-dose: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Week 44 pre-dose | 2.2 (8.9) | -1.6 (6.9) | -0.4 (10.1) | -1.4 (8.2) | 0.7 (9.7)
  Week 44 post dose: number analyzed (Participants) | 36 | 38 | 40 | 33 | 38
  Week 44 post dose | 2.9 (6.9) | -1.7 (8.0) | -0.5 (11.0) | -2.8 (7.7) | -0.2 (10.3)
  Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Week 48 | 2.0 (8.9) | -3.7 (7.8) | -2.5 (10.4) | -4.2 (9.5) | -3.1 (9.5)

11. Secondary Outcome: Changes From Baseline in Body Weight During the Study
Description: Body weight was measured in kilograms.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
  Overall number of participants analyzed include only those for whom body weight was measured and analyzed during the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
kilograms
  Week 12 | 0.14 (3.38) | -0.87 (3.12) | 0.21 (1.78) | -0.38 (1.80) | -0.04 (2.39)
  Week 24: number analyzed (Participants) | 39 | 38 | 41 | 36 | 40
  Week 24 | 0.33 (4.10) | -0.03 (3.48) | -0.07 (2.63) | -0.13 (2.37) | -0.39 (3.73)
  Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Week 36 | 0.32 (5.15) | -0.14 (2.90) | 0.27 (3.42) | 0.15 (2.36) | -0.04 (4.19)
  Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Week 48 | 0.21 (4.42) | 0.45 (3.41) | 0.80 (3.84) | -0.14 (3.32) | 0.11 (4.24)

12. Secondary Outcome: Changes From Baseline in Electrocardiogram (ECG) Intervals During the Study (QTcB, QTcF, PR, QRS, QT, RR)
Description: Electrocardiogram (ECG) intervals (QTcB= QT interval corrected for heart rate (Bazett's formula); QTcF= QT interval corrected for heart rate (Fridericia's formula)) were measured in milliseconds.
Time Frame: Baseline, Week 12 and Week 48
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
  Overall number of participants analyzed include only those for whom electrocardiogram data was measured and analyzed during the study.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 40 | 38 | 42 | 36 | 41
msec
  QTcB Week 12: number analyzed (Participants) | 38 | 36 | 42 | 34 | 40
  QTcB Week 12 | 3.4 (32.7) | -2.8 (29.9) | -5.6 (41.8) | 1.5 (18.2) | -1.9 (31.4)
  QTcB Week 48: number analyzed (Participants) | 35 | 37 | 40 | 31 | 39
  QTcB Week 48 | -2.5 (34.8) | -5.8 (36.5) | -5.9 (22.2) | -4.7 (21.0) | -5.7 (27.7)
  QTcF Week 12: number analyzed (Participants) | 37 | 32 | 35 | 32 | 39
  QTcF Week 12 | 4.5 (27.5) | -2.5 (22.4) | -2.2 (14.2) | -0.5 (17.0) | -3.0 (18.8)
  QTcF Week 48: number analyzed (Participants) | 35 | 32 | 34 | 29 | 38
  QTcF Week 48 | -0.1 (30.7) | -6.1 (31.4) | -0.2 (15.6) | -2.2 (20.0) | 4.6 (44.6)
  PR Week 12: number analyzed (Participants) | 39 | 37 | 42 | 36 | 41
  PR Week 12 | -1.7 (23.3) | -1.0 (23.7) | -19.6 (102.1) | 3.2 (18.2) | -9.5 (32.3)
  PR Week 48: number analyzed (Participants) | 37 | 38 | 40 | 33 | 40
  PR Week 48 | 2.6 (33.7) | 17.5 (128.8) | 4.0 (163.0) | 0.8 (18.9) | -2.8 (26.5)
  QRS Week 12 | 2.6 (22.3) | -2.9 (10.8) | -1.8 (7.6) | -0.2 (5.4) | 6.1 (42.8)
  QRS Week 48: number analyzed (Participants) | 38 | 38 | 40 | 33 | 40
  QRS Week 48 | 5.6 (21.4) | -1.5 (16.1) | -4.0 (13.0) | 0.6 (16.2) | 0.1 (18.7)
  QT Week 12 | -2.0 (46.6) | 1.7 (34.0) | 9.5 (21.4) | 3.8 (25.6) | 11.5 (80.8)
  QT Week 48: number analyzed (Participants) | 38 | 38 | 40 | 33 | 40
  QT Week 48 | -0.7 (33.4) | 3.1 (29.9) | 3.9 (22.8) | 5.4 (26.7) | 0.7 (31.6)
  RR Week 12: number analyzed (Participants) | 39 | 36 | 42 | 34 | 41
  RR Week 12 | 3.3 (99.3) | -22.5 (212.6) | 75.8 (179.3) | 11.0 (125.1) | -17.0 (182.1)
  RR Week 48: number analyzed (Participants) | 37 | 36 | 40 | 31 | 40
  RR Week 48 | -0.6 (116.1) | 11.9 (187.1) | 65.2 (139.0) | 44.3 (124.0) | 25.1 (148.5)

13. Secondary Outcome: Changes From Baseline in Hematology Parameters During the Study (Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils)
Description: Basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils were measured in number of white blood cells per liter (10^9/L).
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44 and Week 48
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: 10^9 white blood cells per liter
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
10^9 white blood cells per liter
  Basophils Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Basophils Week 1 | 0.000 (0.0387) | 0.000 (0.0329) | -0.002 (0.0408) | 0.007 (0.0264) | 0.008 (0.0350)
  Basophils Week 2: number analyzed (Participants) | 42 | 38 | 43 | 41 | 41
  Basophils Week 2 | 0.002 (0.0269) | 0.003 (0.0283) | 0.000 (0.0488) | 0.000 (0.0316) | 0.005 (0.0384)
  Basophils Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Basophils Week 4 | 0.002 (0.0474) | 0.005 (0.0324) | -0.007 (0.0463) | 0.005 (0.0312) | 0.005 (0.0312)
  Basophils Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Basophils Week 8 | -0.002 (0.0353) | 0.000 (0.0229) | -0.005 (0.0384) | 0.003 (0.0367) | 0.002 (0.0418)
  Basophils Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Basophils Week 12 | 0.002 (0.0353) | 0.003 (0.0280) | -0.002 (0.0462) | 0.000 (0.0329) | 0.010 (0.0374)
  Basophils Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Basophils Week 16 | 0.010 (0.0431) | 0.005 (0.0324) | -0.007 (0.0463) | 0.000 (0.0329) | 0.008 (0.0417)
  Basophils Week 20: number analyzed (Participants) | 39 | 39 | 41 | 37 | 39
  Basophils Week 20 | -0.003 (0.0362) | 0.003 (0.0362) | 0.000 (0.0500) | 0.005 (0.0329) | 0.000 (0.0397)
  Basophils Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Basophils Week 24 | 0.000 (0.0397) | 0.005 (0.0324) | -0.003 (0.0530) | 0.008 (0.0368) | 0.005 (0.0389)
  Basophils Week 28: number analyzed (Participants) | 39 | 38 | 40 | 35 | 40
  Basophils Week 28 | 0.005 (0.0394) | 0.000 (0.0329) | 0.008 (0.0526) | 0.011 (0.0323) | 0.005 (0.0450)
  Basophils Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Basophils Week 32 | 0.000 (0.0324) | 0.005 (0.0320) | -0.010 (0.0441) | 0.009 (0.0379) | 0.010 (0.0384)
  Basophils Week 36: number analyzed (Participants) | 37 | 38 | 41 | 33 | 39
  Basophils Week 36 | 0.000 (0.0408) | 0.003 (0.0283) | -0.002 (0.0474) | 0.012 (0.0415) | 0.013 (0.0409)
  Basophils Week 40: number analyzed (Participants) | 36 | 38 | 40 | 34 | 38
  Basophils Week 40 | 0.003 (0.0506) | 0.005 (0.0399) | -0.010 (0.0379) | 0.006 (0.0343) | 0.000 (0.0403)
  Basophils Week 44: number analyzed (Participants) | 36 | 37 | 41 | 34 | 36
  Basophils Week 44 | 0.006 (0.0410) | 0.003 (0.0372) | 0.000 (0.0387) | 0.006 (0.0422) | 0.000 (0.0338)
  Basophils Week 48: number analyzed (Participants) | 38 | 36 | 40 | 32 | 39
  Basophils Week 48 | -0.005 (0.0462) | 0.003 (0.291) | -0.010 (0.0441) | 0.006 (0.0354) | 0.000 (0.0324)
  Eosinophils Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Eosinophils Week 1 | 0.010 (0.0860) | 0.016 (0.0718) | -0.002 (0.0801) | -0.005 (0.0999) | 0.017 (0.0636)
  Eosinophils Week 2: number analyzed (Participants) | 42 | 38 | 43 | 41 | 41
  Eosinophils Week 2 | 0.005 (0.0731) | 0.013 (0.0777) | 0.002 (0.0913) | 0.002 (0.0880) | 0.029 (0.0929)
  Eosinophils Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Eosinophils Week 4 | 0.002 (0.0987) | 0.016 (0.0594) | 0.002 (0.0780) | 0.005 (0.0999) | 0.027 (0.0895)
  Eosinophils Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Eosinophils Week 8 | 0.024 (0.0969) | -0.003 (0.0707) | 0.000 (0.1000) | 0.008 (0.0941) | 0.005 (0.0669)
  Eosinophils Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Eosinophils Week 12 | 0.020 (0.0954) | 0.010 (0.0882) | 0.002 (0.0831) | -0.026 (0.1155) | 0.017 (0.0704)
  Eosinophils Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Eosinophils Week 16 | 0.045 (0.1253) | 0.021 (0.0935) | 0.010 (0.0759) | -0.005 (0.1559) | 0.033 (0.0829)
  Eosinophils Week 20: number analyzed (Participants) | 39 | 39 | 41 | 37 | 39
  Eosinophils Week 20 | 0.036 (0.1038) | 0.026 (0.1186) | 0.024 (0.1157) | -0.014 (0.1228) | 0.038 (0.0935)
  Eosinophils Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Eosinophils Week 24 | 0.031 (0.1301) | 0.013 (0.0844) | 0.058 (0.2111) | -0.019 (0.1238) | 0.037 (0.1192)
  Eosinophils Week 28: number analyzed (Participants) | 39 | 38 | 40 | 35 | 40
  Eosinophils Week 28 | 0.036 (0.0986) | 0.018 (0.0926) | 0.053 (0.1826) | -0.000 (0.1213) | 0.025 (0.0870)
  Eosinophils Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Eosinophils Week 32 | 0.049 (0.1502) | 0.033 (0.0838) | 0.020 (0.1418) | 0.024 (0.1577) | 0.041 (0.1141)
  Eosinophils Week 36: number analyzed (Participants) | 37 | 38 | 41 | 33 | 39
  Eosinophils Week 36 | 0.054 (0.1726) | 0.018 (0.0955) | 0.022 (0.0909) | 0.027 (0.1526) | 0.015 (0.0961)
  Eosinophils Week 40: number analyzed (Participants) | 36 | 38 | 40 | 34 | 38
  Eosinophils Week 40 | 0.050 (0.1444) | 0.018 (0.0865) | 0.018 (0.0958) | 0.015 (0.1971) | 0.039 (0.1128)
  Eosinophils Week 44: number analyzed (Participants) | 36 | 37 | 41 | 34 | 36
  Eosinophils Week 44 | 0.072 (0.1523) | 0.019 (0.0908) | 0.024 (0.0994) | -0.009 (0.1798) | 0.006 (0.0893)
  Eosinophils Week 48: number analyzed (Participants) | 38 | 36 | 40 | 32 | 39
  Eosinophils Week 48 | 0.045 (0.1811) | 0.006 (0.0754) | 0.023 (0.0891) | 0.009 (0.2833) | -0.005 (0.0857)
  Leukocytes Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Leukocytes Week 1 | -0.271 (1.1885) | -0.597 (1.1490) | -0.656 (1.2593) | -1.029 (1.6496) | -0.285 (1.6896)
  Leukocytes Week 2 | 0.157 (1.3195) | -0.131 (2.1769) | -0.309 (1.3735) | -0.954 (2.0441) | -0.322 (1.5501)
  Leukocytes Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Leukocytes Week 4 | -0.049 (1.1938) | -0.411 (1.1988) | -0.336 (1.5088) | -1.017 (1.9397) | -0.656 (1.4264)
  Leukocytes Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Leukocytes Week 8 | 0.429 (1.7036) | -0.333 (1.4014) | -0.185 (1.2889) | -1.071 (1.9639) | -0.629 (1.5489)
  Leukocytes Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Leukocytes Week 12 | 0.190 (1.6223) | -0.438 (1.3854) | -0.495 (1.6904) | -0.997 (2.1806) | -0.634 (1.6084)
  Leukocytes Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Leukocytes Week 16 | -0.400 (1.5616) | -0.839 (1.8179) | -0.590 (1.4668) | -1.318 (2.3324) | -0.293 (1.8427)
  Leukocytes Week 20: number analyzed (Participants) | 39 | 39 | 41 | 37 | 40
  Leukocytes Week 20 | -0.936 (1.2756) | -1.100 (1.5599) | -0.432 (1.3032) | -0.932 (2.2832) | -0.455 (1.7116)
  Leukocytes Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Leukocytes Week 24 | -1.251 (1.3888) | -0.884 (1.7768) | -0.495 (1.4216) | -1.119 (2.2807) | -0.765 (1.8691)
  Leukocytes Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Leukocytes Week 28 | -0.700 (1.8180) | -0.316 (2.3086) | -0.100 (1.4942) | -0.894 (1.7119) | -0.342 (1.5683)
  Leukocytes Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Leukocytes Week 32 | -0.762 (1.4273) | -0.862 (2.0091) | -0.330 (1.5750) | -0.918 (2.6184) | -0.505 (1.4800)
  Leukocytes Week 36: number analyzed (Participants) | 37 | 38 | 41 | 33 | 39
  Leukocytes Week 36 | -0.541 (1.5971) | -0.974 (1.7389) | -0.366 (1.4549) | -1.082 (2.3389) | -0.126 (2.2565)
  Leukocytes Week 40: number analyzed (Participants) | 36 | 38 | 41 | 34 | 38
  Leukocytes Week 40 | -0.783 (1.7693) | -0.826 (1.5942) | -0.437 (1.7878) | -1.226 (2.3856) | -0.266 (1.7976)
  Leukocytes Week 44: number analyzed (Participants) | 37 | 37 | 41 | 34 | 36
  Leukocytes Week 44 | -1.065 (1.6070) | -0.978 (1.8151) | -0.537 (1.5641) | -1.032 (2.1585) | -0.825 (1.8917)
  Leukocytes Week 48: number analyzed (Participants) | 38 | 36 | 40 | 32 | 39
  Leukocytes Week 48 | -0.739 (1.7774) | -0.869 (1.7109) | -0.473 (1.7104) | -1.225 (2.5952) | -0.777 (1.8593)
  Lymphocytes Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Lymphocytes Week 1 | -0.083 (0.5074) | -0.024 (0.4142) | 0.044 (0.5039) | -0.017 (0.4189) | 0.020 (0.3006)
  Lymphocytes Week 2: number analyzed (Participants) | 42 | 38 | 43 | 41 | 41
  Lymphocytes Week 2 | 0.105 (0.3246) | 0.026 (0.4137) | 0.021 (0.6006) | 0.007 (0.3643) | 0.161 (0.4277)
  Lymphocytes Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Lymphocytes Week 4 | 0.037 (0.4386) | 0.024 (0.3259) | 0.010 (0.6003) | -0.032 (0.3996) | 0.095 (0.3263)
  Lymphocytes Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Lymphocytes Week 8 | 0.120 (0.3776) | 0.054 (0.3783) | 0.063 (0.5928) | 0.053 (0.4980) | 0.129 (0.3939)
  Lymphocytes Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Lymphocytes Week 12 | 0.041 (0.3647) | 0.051 (0.4167) | 0.000 (0.5640) | -0.047 (0.3703) | 0.061 (0.3301)
  Lymphocytes Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Lymphocytes Week 16 | 0.052 (0.5567) | 0.071 (0.3571) | 0.026 (0.5539) | -0.029 (0.4991) | 0.135 (0.4197)
  Lymphocytes Week 20: number analyzed (Participants) | 39 | 39 | 41 | 37 | 39
  Lymphocytes Week 20 | 0.003 (0.4934) | 0.008 (0.3970) | 0.149 (0.4675) | -0.035 (0.4566) | 0.126 (0.4216)
  Lymphocytes Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Lymphocytes Week 24 | -0.041 (0.3905) | 0.050 (0.3630) | 0.048 (0.4455) | -0.036 (0.3788) | 0.053 (0.3974)
  Lymphocytes Week 28: number analyzed (Participants) | 39 | 38 | 40 | 35 | 40
  Lymphocytes Week 28 | 0.036 (0.5869) | 0.105 (0.3594) | 0.210 (0.5999) | 0.103 (0.5544) | 0.172 (0.3776)
  Lymphocytes Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Lymphocytes Week 32 | -0.000 (0.5109) | 0.103 (0.4233) | 0.083 (0.6524) | 0.112 (0.5056) | 0.146 (0.3966)
  Lymphocytes Week 36: number analyzed (Participants) | 37 | 38 | 41 | 33 | 39
  Lymphocytes Week 36 | 0.078 (0.4894) | 0.039 (0.4227) | 0.134 (0.5673) | 0.103 (0.5491) | 0.118 (0.3810)
  Lymphocytes Week 40: number analyzed (Participants) | 36 | 38 | 40 | 34 | 38
  Lymphocytes Week 40 | 0.139 (0.4871) | 0.168 (0.4281) | 0.120 (0.6018) | 0.038 (0.4335) | 0.176 (0.3709)
  Lymphocytes Week 44: number analyzed (Participants) | 36 | 37 | 41 | 34 | 36
  Lymphocytes Week 44 | -0.008 (0.5390) | 0.105 (0.4136) | 0.124 (0.5366) | 0.115 (0.4881) | 0.153 (0.4462)
  Lymphocytes Week 48: number analyzed (Participants) | 38 | 36 | 40 | 32 | 39
  Lymphocytes Week 48 | 0.066 (0.5313) | 0.103 (0.3645) | 0.078 (0.5041) | 0.019 (0.3763) | 0.072 (0.3755)
  Monocytes Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Monocytes Week 1 | 0.007 (0.2184) | -0.008 (0.1477) | -0.012 (0.1679) | -0.088 (0.2315) | -0.027 (0.1724)
  Monocytes Week 2: number analyzed (Participants) | 42 | 38 | 43 | 41 | 41
  Monocytes Week 2 | 0.076 (0.1358) | -0.011 (0.1673) | 0.014 (0.1897) | -0.095 (0.2701) | -0.010 (0.1882)
  Monocytes Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Monocytes Week 4 | 0.032 (0.1588) | -0.021 (0.1473) | -0.040 (0.1862) | -0.066 (0.2404) | -0.085 (0.1459)
  Monocytes Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Monocytes Week 8 | 0.059 (0.1910) | -0.041 (0.1743) | 0.005 (0.1580) | -0.103 (0.2520) | -0.071 (0.1834)
  Monocytes Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Monocytes Week 12 | 0.020 (0.1913) | -0.031 (0.1608) | -0.033 (0.1686) | -0.105 (0.2630) | -0.059 (0.1414)
  Monocytes Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Monocytes Week 16 | -0.007 (0.1629) | -0.050 (0.1673) | -0.024 (0.1265) | -0.079 (0.2384) | -0.043 (0.1752)
  Monocytes Week 20: number analyzed (Participants) | 39 | 39 | 41 | 37 | 39
  Monocytes Week 20 | -0.008 (0.1783) | -0.041 (0.1534) | -0.015 (0.1509) | -0.081 (0.2448) | -0.003 (0.1899)
  Monocytes Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Monocytes Week 24 | -0.026 (0.1292) | -0.034 (0.1361) | 0.003 (0.1476) | -0.056 (0.2602) | -0.027 (0.1921)
  Monocytes Week 28: number analyzed (Participants) | 39 | 38 | 40 | 35 | 40
  Monocytes Week 28 | 0.026 (0.2087) | 0.042 (0.1981) | 0.055 (0.1724) | -0.029 (0.2729) | -0.012 (0.1911)
  Monocytes Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Monocytes Week 32 | 0.064 (0.2356) | -0.005 (0.1731) | -0.003 (0.1271) | -0.035 (0.2684) | 0.010 (0.1744)
  Monocytes Week 36: number analyzed (Participants) | 37 | 38 | 41 | 33 | 39
  Monocytes Week 36 | 0.054 (0.1626) | -0.024 (0.1792) | 0.032 (0.1404) | -0.036 (0.2644) | 0.049 (0.2327)
  Monocytes Week 40: number analyzed (Participants) | 36 | 38 | 40 | 34 | 38
  Monocytes Week 40 | 0.053 (0.1647) | 0.008 (0.1323) | 0.020 (0.1636) | -0.059 (0.2830) | -0.018 (0.1504)
  Monocytes Week 44: number analyzed (Participants) | 36 | 37 | 41 | 34 | 36
  Monocytes Week 44 | 0.019 (0.1939) | -0.008 (0.1588) | 0.044 (0.1644) | -0.032 (0.2446) | -0.019 (0.2202)
  Monocytes Week 48: number analyzed (Participants) | 38 | 36 | 40 | 32 | 39
  Monocytes Week 48 | 0.021 (0.2145) | 0.000 (0.1707) | -0.013 (0.1399) | -0.078 (0.2511) | -0.077 (0.1709)
  Neutrophils Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Neutrophils Week 1 | -0.200 (1.0959) | -0.558 (0.9627) | -0.693 (1.2971) | -0.934 (1.4768) | -0.325 (1.5720)
  Neutrophils Week 2: number analyzed (Participants) | 42 | 38 | 43 | 41 | 41
  Neutrophils Week 2 | -0.026 (1.1945) | -0.418 (1.1627) | -0.337 (1.3109) | -0.880 (1.8457) | -0.537 (1.3989)
  Neutrophils Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Neutrophils Week 4 | -0.102 (1.0044) | -0.405 (1.1246) | -0.290 (1.3463) | -0.924 (1.9975) | -0.732 (1.4028)
  Neutrophils Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Neutrophils Week 8 | 0.249 (1.5358) | -0.346 (1.2640) | -0.256 (1.3898) | -1.021 (1.7129) | -0.717 (1.4589)
  Neutrophils Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Neutrophils Week 12 | 0.117 (1.5103) | -0.456 (1.1227) | -0.458 (1.6879) | -0.832 (2.2192) | -0.673 (1.3887)
  Neutrophils Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Neutrophils Week 16 | -0.490 (1.6866) | -0.879 (1.5752) | -0.617 (1.6027) | -1.203 (2.2840) | -0.448 (1.6816)
  Neutrophils Week 20: number analyzed (Participants) | 39 | 39 | 41 | 37 | 39
  Neutrophils Week 20 | -0.972 (1.2085) | -1.069 (1.4219) | -0.595 (1.4319) | -0.827 (2.2663) | -0.618 (1.5716)
  Neutrophils Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Neutrophils Week 24 | -1.210 (1.4067) | -0.895 (1.6288) | -0.593 (1.5309) | -1.011 (2.2968) | -0.850 (1.6461)
  Neutrophils Week 28: number analyzed (Participants) | 39 | 38 | 40 | 35 | 40
  Neutrophils Week 28 | -0.774 (1.8189) | -0.484 (2.2620) | -0.555 (1.2608) | -0.949 (1.7676) | -0.568 (1.3889)
  Neutrophils Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Neutrophils Week 32 | -0.869 (1.2796) | -0.969 (1.8241) | -0.433 (1.7889) | -1.038 (2.4800) | -0.718 (1.4299)
  Neutrophils Week 36: number analyzed (Participants) | 37 | 38 | 41 | 33 | 39
  Neutrophils Week 36 | -0.722 (1.6422) | -0.992 (1.6583) | -0.541 (1.5519) | -1.185 (2.1881) | -0.354 (2.1441)
  Neutrophils Week 40: number analyzed (Participants) | 36 | 38 | 40 | 34 | 38
  Neutrophils Week 40 | -1.006 (1.7393) | -0.992 (1.4740) | -0.575 (1.9567) | -1.229 (2.4065) | -0.495 (1.5857)
  Neutrophils Week 44: number analyzed (Participants) | 36 | 37 | 41 | 34 | 36
  Neutrophils Week 44 | -0.978 (1.2444) | -1.086 (1.6049) | -0.717 (1.6966) | -1.109 (2.2673) | -0.983 (1.6556)
  Neutrophils Week 48: number analyzed (Participants) | 38 | 36 | 40 | 32 | 39
  Neutrophils Week 48 | -0.861 (1.6858) | -0.939 (1.5670) | -0.558 (1.7944) | -1.178 (2.6503) | -0.805 (1.6631)

14. Secondary Outcome: Changes From Baseline in Hematology Parameters During the Study (Erythrocytes Mean Corpuscular Hemoglobin (HGB) Concentration, Hemoglobin)
Description: Erythrocytes mean corpuscular hemoglobin (HGB) concentration and hemoglobin were measured in grams per liter (g/L).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
g/L
  Ery. mean corpuscular HGB Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Ery. mean corpuscular HGB Week 1 | -2.293 (8.4594) | 0.789 (8.9719) | -1.860 (8.0551) | 0.927 (9.1088) | 1.200 (12.2395)
  Ery. mean corpuscular HGB Week 2 | -2.310 (7.9923) | 2.564 (9.8216) | 0.465 (8.4778) | 0.707 (8.6263) | 2.854 (10.1822)
  Ery. mean corpuscular HGB Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Ery. mean corpuscular HGB Week 4 | -3.927 (10.0633) | 1.474 (10.5849) | -2.500 (11.5045) | -0.878 (9.4026) | 1.756 (11.8697)
  Ery. mean corpuscular HGB Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Ery. mean corpuscular HGB Week 8 | -5.195 (11.7158) | -1.897 (11.3249) | -3.780 (10.7576) | -3.079 (10.7033) | 0.610 (12.7493)
  Ery. mean corpuscular HGB Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Ery. mean corpuscular HGB Week 12 | -7.927 (14.6704) | -3.179 (13.4122) | -3.907 (11.5404) | -2.684 (9.4099) | 1.732 (13.3959)
  Ery. mean corpuscular HGB Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Ery. mean corpuscular HGB Week 16 | -6.286 (12.3393) | -3.000 (14.5751) | -5.262 (12.1917) | -1.026 (11.6816) | -0.700 (16.1026)
  Ery. mean corpuscular HGB Week 20: number analyzed (Participants) | 40 | 39 | 41 | 37 | 40
  Ery. mean corpuscular HGB Week 20 | -5.050 (12.8102) | 0.923 (11.8108) | -1.902 (12.8078) | 0.919 (8.7349) | 0.200 (16.1725)
  Ery. mean corpuscular HGB Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Ery. mean corpuscular HGB Week 24 | 1.000 (10.9232) | 4.132 (10.3849) | -0.625 (14.6685) | 4.583 (11.3121) | 4.250 (13.4064)
  Ery. mean corpuscular HGB Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Ery. mean corpuscular HGB Week 28 | 2.179 (10.3285) | 4.658 (9.6906) | 1.707 (9.9505) | 4.400 (13.7524) | 6.150 (12.5382)
  Ery. mean corpuscular HGB Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Ery. mean corpuscular HGB Week 32 | 6.308 (9.7796) | 10.231 (9.5957) | 4.850 (11.3692) | 7.971 (12.3497) | 10.462 (12.9855)
  Ery. mean corpuscular HGB Week 36: number analyzed (Participants) | 38 | 38 | 41 | 33 | 39
  Ery. mean corpuscular HGB Week 36 | 5.500 (9.7779) | 10.921 (10.2229) | 2.732 (12.4097) | 6.788 (12.2034) | 9.462 (12.7998)
  Ery. mean corpuscular HGB Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 38
  Ery. mean corpuscular HGB Week 40 | 3.108 (9.8736) | 8.237 (12.0706) | 4.976 (11.5639) | 9.088 (11.5480) | 9.079 (11.5393)
  Ery. mean corpuscular HGB Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 36
  Ery. mean corpuscular HGB Week 44 | 6.297 (10.6975) | 7.289 (12.6254) | 3.415 (12.6293) | 6.353 (14.3038) | 9.278 (12.8076)
  Ery. mean corpuscular HGB Week 48: number analyzed (Participants) | 38 | 37 | 41 | 33 | 40
  Ery. mean corpuscular HGB Week 48 | 5.079 (10.4916) | 7.216 (9.3812) | 2.122 (11.8769) | 5.394 (12.9300) | 8.250 (11.3448)
  Hemoglobin Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Hemoglobin Week 1 | -4.854 (5.6726) | 0.000 (5.6569) | 1.302 (5.1480) | 0.512 (6.0462) | -0.875 (4.8368)
  Hemoglobin Week 2 | -4.810 (6.5154) | -0.359 (5.2339) | 0.070 (6.5915) | -1.561 (6.7047) | 0.317 (5.3499)
  Hemoglobin Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Hemoglobin Week 4 | -4.390 (7.5162) | 0.895 (7.6434) | 0.881 (6.4551) | 0.512 (5.7189) | 1.195 (5.8916)
  Hemoglobin Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Hemoglobin Week 8 | -4.561 (7.0995) | 0.308 (7.0865) | 2.195 (7.7628) | 0.553 (6.8010) | 1.195 (7.4439)
  Hemoglobin Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Hemoglobin Week 12 | -5.220 (6.7879) | 0.692 (7.7601) | 2.488 (7.6512) | 0.868 (7.3344) | 2.488 (8.2344)
  Hemoglobin Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Hemoglobin Week 16 | -1.619 (6.4768) | 2.579 (8.3880) | 1.524 (8.7853) | 1.737 (7.3547) | 3.125 (7.7400)
  Hemoglobin Week 20: number analyzed (Participants) | 40 | 39 | 41 | 37 | 40
  Hemoglobin Week 20 | -0.400 (7.3233) | 2.667 (8.6764) | 2.268 (6.9822) | 1.892 (7.6186) | 2.925 (7.7207)
  Hemoglobin Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Hemoglobin Week 24 | 0.564 (8.1879) | 3.658 (9.0622) | 4.075 (8.0714) | 2.000 (6.6462) | 3.425 (6.2834)
  Hemoglobin Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Hemoglobin Week 28 | -1.513 (8.0259) | 3.342 (8.9511) | 3.122 (8.6261) | 0.857 (7.2645) | 3.400 (8.6730)
  Hemoglobin Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Hemoglobin Week 32 | -0.282 (8.2684) | 4.487 (8.3094) | 4.300 (9.4032) | 2.118 (7.4254) | 5.615 (8.6378)
  Hemoglobin Week 36: number analyzed (Participants) | 38 | 38 | 41 | 33 | 39
  Hemoglobin Week 36 | 0.947 (9.1738) | 6.053 (8.1405) | 4.293 (9.5766) | 3.818 (7.3334) | 4.949 (8.4851)
  Hemoglobin Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 38
  Hemoglobin Week 40 | 1.432 (9.1090) | 5.868 (8.7863) | 4.317 (9.6552) | 3.618 (7.8277) | 4.132 (7.7987)
  Hemoglobin Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 36
  Hemoglobin Week 44 | 1.486 (10.1040) | 5.000 (9.2998) | 3.659 (9.1750) | 4.912 (8.5895) | 4.722 (8.5511)
  Hemoglobin Week 48: number analyzed (Participants) | 38 | 37 | 41 | 33 | 40
  Hemoglobin Week 48 | 2.474 (9.7002) | 5.270 (9.1974) | 3.780 (9.9210) | 4.030 (9.2550) | 4.725 (7.3554)

15. Secondary Outcome: Changes From Baseline in Hematology Parameters During the Study (Erythrocytes Mean Corpuscular Hemoglobin (HGB))
Description: Erythrocytes mean corpuscular hemoglobin (HGB) was measured in picograms (pg).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
picograms (pg)
  Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Week 1 | -0.073 (0.4980) | 0.058 (0.4624) | -0.049 (0.4050) | 0.073 (0.3975) | -0.055 (0.4455)
  Week 2 | -0.050 (0.3890) | 0.126 (0.5149) | 0.023 (0.4225) | 0.066 (0.4357) | 0.085 (0.4287)
  Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Week 4 | -0.112 (0.5501) | 0.089 (0.5584) | 0.060 (0.5910) | 0.012 (0.4691) | 0.066 (0.6085)
  Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Week 8 | -0.110 (0.6778) | 0.141 (0.6801) | 0.007 (0.5926) | 0.034 (0.6851) | 0.095 (0.7994)
  Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Week 12 | -0.285 (0.6770) | 0.023 (0.7253) | 0.091 (0.8358) | -0.132 (0.8335) | 0.039 (1.0454)
  Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Week 16 | -0.233 (0.7281) | 0.097 (0.8824) | 0.014 (0.9236) | -0.118 (0.8440) | -0.067 (1.1713)
  Week 20: number analyzed (Participants) | 40 | 39 | 41 | 37 | 40
  Week 20 | -0.290 (0.8145) | -0.033 (0.9172) | 0.029 (0.9819) | -0.035 (0.7013) | 0.075 (1.0824)
  Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Week 24 | -0.249 (1.0443) | 0.108 (0.9947) | -0.057 (1.1804) | -0.097 (0.7284) | -0.007 (1.2338)
  Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Week 28 | -0.103 (1.0101) | 0.029 (0.7241) | -0.122 (1.1130) | -0.211 (0.8277) | 0.020 (1.2950)
  Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Week 32 | 0.003 (1.2619) | 0.297 (0.8561) | 0.058 (1.1522) | 0.026 (0.7684) | 0.167 (1.2472)
  Week 36: number analyzed (Participants) | 38 | 38 | 41 | 33 | 39
  Week 36 | -0.082 (1.3242) | 0.237 (0.8722) | -0.093 (1.0792) | -0.248 (0.8581) | 0.118 (1.1473)
  Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 38
  Week 40 | -0.170 (1.3453) | 0.134 (0.8960) | -0.134 (1.2095) | -0.147 (0.8645) | 0.034 (1.0839)
  Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 36
  Week 44 | 0.097 (1.3103) | 0.129 (0.8742) | -0.080 (1.1771) | -0.159 (0.7480) | 0.108 (1.2532)
  Week 48: number analyzed (Participants) | 38 | 37 | 41 | 33 | 40
  Week 48 | 0.137 (1.4139) | 0.178 (0.9369) | -0.120 (1.1279) | -0.030 (0.7888) | 0.140 (1.2161)

16. Secondary Outcome: Changes From Baseline in Hematology Parameters During the Study (Erythrocytes Mean Corpuscular Volume)
Description: Erythrocytes mean corpuscular volume was measured in femtolitres (fL).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: femtolitres (fL)
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
femtolitres (fL)
  Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Week 1 | 0.422 (1.8855) | -0.087 (1.9540) | 0.386 (2.2542) | -0.017 (2.1066) | -0.510 (2.7686)
  Week 2 | 0.450 (1.8867) | -0.362 (2.1689) | -0.021 (1.8767) | -0.039 (2.3876) | -0.549 (2.5751)
  Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Week 4 | 0.829 (2.3409) | -0.163 (2.4631) | 0.945 (3.2325) | 0.354 (2.8851) | -0.259 (2.5328)
  Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Week 8 | 1.163 (3.6524) | 0.938 (2.9445) | 1.110 (3.0283) | 0.916 (3.0058) | 0.090 (3.5125)
  Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Week 12 | 1.478 (3.9560) | 0.951 (3.4617) | 1.367 (3.8471) | 0.342 (3.1129) | -0.390 (3.3907)
  Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Week 16 | 1.107 (3.4022) | 1.168 (3.7760) | 1.571 (4.3326) | -0.016 (3.6944) | 0.048 (4.4345)
  Week 20: number analyzed (Participants) | 40 | 39 | 41 | 37 | 40
  Week 20 | 0.497 (3.5197) | -0.349 (2.8975) | 0.649 (3.7758) | -0.338 (2.5959) | 0.202 (4.2993)
  Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Week 24 | -1.033 (2.9007) | -0.858 (2.1793) | 0.143 (4.9985) | -1.522 (3.1692) | -1.195 (3.5759)
  Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Week 28 | -0.910 (2.6477) | -1.184 (2.3264) | -0.754 (3.3662) | -1.854 (3.6605) | -1.638 (3.3447)
  Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Week 32 | -1.654 (2.7565) | -1.851 (2.4024) | -1.075 (3.5390) | -2.071 (3.7652) | -2.351 (3.1052)
  Week 36: number analyzed (Participants) | 38 | 38 | 41 | 33 | 39
  Week 36 | -1.724 (3.1037) | -2.266 (2.3516) | -0.912 (3.9627) | -2.558 (3.8468) | -2.236 (3.2869)
  Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 38
  Week 40 | -1.386 (2.8575) | -1.882 (3.1285) | -1.698 (3.0263) | -2.885 (3.1443) | -2.421 (2.9445)
  Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 36
  Week 44 | -1.405 (3.4627) | -1.632 (3.4207) | -1.117 (3.4616) | -2.171 (4.4367) | -2.186 (3.4915)
  Week 48: number analyzed (Participants) | 38 | 37 | 41 | 33 | 40
  Week 48 | -0.942 (3.5913) | -1.492 (2.5065) | -0.846 (3.1243) | -1.527 (3.6540) | -1.788 (3.5554)

17. Secondary Outcome: Changes From Baseline in Hematology Parameters During the Study (Erythrocytes)
Description: Erythrocytes was measured in number of red blood cells per liter (10^12/L).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: 10^12 red blood cells per liter
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
10^12 red blood cells per liter
  Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Week 1 | -0.148 (0.2071) | -0.008 (0.1927) | 0.050 (0.1773) | 0.008 (0.2109) | -0.017 (0.1609)
  Week 2 | -0.149 (0.2244) | -0.029 (0.1788) | -0.004 (0.2280) | -0.063 (0.2236) | 0.000 (0.1809)
  Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Week 4 | -0.132 (0.2780) | 0.018 (0.2535) | 0.023 (0.2135) | 0.013 (0.1955) | 0.031 (0.2065)
  Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Week 8 | -0.135 (0.2546) | -0.011 (0.2206) | 0.074 (0.2466) | 0.014 (0.2190) | 0.026 (0.2264)
  Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Week 12 | -0.131 (0.2678) | 0.021 (0.2561) | 0.069 (0.2419) | 0.051 (0.2243) | 0.075 (0.2393)
  Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Week 16 | -0.020 (0.2375) | 0.075 (0.2898) | 0.047 (0.2810) | 0.074 (0.2255) | 0.110 (0.2533)
  Week 20: number analyzed (Participants) | 40 | 39 | 41 | 37 | 40
  Week 20 | 0.036 (0.2618) | 0.096 (0.2855) | 0.068 (0.2089) | 0.064 (0.2273) | 0.081 (0.2191)
  Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Week 24 | 0.059 (0.2639) | 0.110 (0.2974) | 0.142 (0.2573) | 0.074 (0.2250) | 0.110 (0.1931)
  Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Week 28 | -0.034 (0.2453) | 0.108 (0.2681) | 0.122 (0.2445) | 0.058 (0.2359) | 0.106 (0.2567)
  Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Week 32 | -0.010 (0.2461) | 0.104 (0.2660) | 0.133 (0.2716) | 0.061 (0.2555) | 0.156 (0.2714)
  Week 36: number analyzed (Participants) | 38 | 38 | 41 | 33 | 39
  Week 36 | 0.044 (0.2524) | 0.166 (0.2542) | 0.156 (0.2849) | 0.161 (0.2399) | 0.145 (0.2377)
  Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 38
  Week 40 | 0.079 (0.2682) | 0.177 (0.2733) | 0.163 (0.2736) | 0.141 (0.2535) | 0.129 (0.2403)
  Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 36
  Week 44 | 0.035 (0.2645) | 0.146 (0.2846) | 0.133 (0.2622) | 0.188 (0.2933) | 0.135 (0.2128)
  Week 48: number analyzed (Participants) | 38 | 37 | 41 | 33 | 40
  Week 48 | 0.061 (0.2693) | 0.146 (0.2994) | 0.141 (0.2747) | 0.135 (0.2934) | 0.129 (0.2354)

18. Secondary Outcome: Changes From Baseline in Hematology Parameters During the Study (Hematocrit)
Description: Hematocrit was measured in volume percentage (%) of red blood cells in blood.
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: volume % of red blood cells
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
volume % of red blood cells
  Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Week 1 | -0.011 (0.0189) | -0.001 (0.0211) | 0.007 (0.0181) | 0.000 (0.0206) | -0.004 (0.0206)
  Week 2 | -0.011 (0.0230) | -0.004 (0.0204) | -0.000 (0.0205) | -0.006 (0.0220) | -0.003 (0.0174)
  Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Week 4 | -0.008 (0.0254) | 0.001 (0.0211) | 0.006 (0.0220) | 0.003 (0.0190) | 0.001 (0.0209)
  Week 8: number analyzed (Participants) | 41 | 39 | 41 | 38 | 41
  Week 8 | -0.007 (0.0239) | 0.003 (0.0244) | 0.012 (0.0237) | 0.005 (0.0208) | 0.003 (0.0232)
  Week 12: number analyzed (Participants) | 41 | 39 | 43 | 38 | 41
  Week 12 | -0.005 (0.0287) | 0.007 (0.0281) | 0.013 (0.0276) | 0.006 (0.0219) | 0.005 (0.0231)
  Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Week 16 | 0.004 (0.0202) | 0.012 (0.0259) | 0.011 (0.0254) | 0.006 (0.0240) | 0.010 (0.0252)
  Week 20: number analyzed (Participants) | 40 | 39 | 41 | 37 | 40
  Week 20 | 0.006 (0.0217) | 0.007 (0.0270) | 0.010 (0.0211) | 0.004 (0.0241) | 0.008 (0.0246)
  Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Week 24 | 0.001 (0.0192) | 0.006 (0.0253) | 0.014 (0.0256) | -0.000 (0.0222) | 0.005 (0.0219)
  Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Week 28 | -0.007 (0.0210) | 0.004 (0.0248) | 0.008 (0.0241) | -0.003 (0.0229) | 0.002 (0.0238)
  Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Week 32 | -0.009 (0.0207) | 0.000 (0.0249) | 0.007 (0.0225) | -0.004 (0.0196) | 0.003 (0.0248)
  Week 36: number analyzed (Participants) | 38 | 38 | 41 | 33 | 39
  Week 36 | -0.004 (0.0222) | 0.004 (0.0228) | 0.009 (0.0258) | 0.003 (0.0221) | 0.003 (0.0234)
  Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 38
  Week 40 | 0.000 (0.0231) | 0.007 (0.0278) | 0.007 (0.0246) | -0.001 (0.0221) | 0.000 (0.0206)
  Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 36
  Week 44 | -0.003 (0.0272) | 0.006 (0.0297) | 0.007 (0.0239) | 0.007 (0.0246) | 0.002 (0.0194)
  Week 48: number analyzed (Participants) | 38 | 37 | 41 | 33 | 40
  Week 48 | 0.001 (0.0243) | 0.007 (0.0257) | 0.009 (0.0260) | 0.005 (0.0252) | 0.004 (0.0212)

19. Secondary Outcome: Changes From Baseline in Hematology Parameters During the Study (Platelets)
Description: Platelets was measured in number of platelets per liter (10^9/L).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
10^9 platelets per liter
  Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Week 1 | -5.073 (30.2609) | -3.368 (25.9515) | 3.209 (30.5883) | -2.098 (24.6412) | -9.325 (23.4109)
  Week 2: number analyzed (Participants) | 42 | 39 | 42 | 41 | 41
  Week 2 | 4.000 (27.3112) | -5.179 (38.2800) | -3.810 (41.8250) | -15.122 (32.8414) | -15.415 (31.7025)
  Week 4: number analyzed (Participants) | 41 | 38 | 41 | 41 | 41
  Week 4 | -3.927 (29.6643) | -6.868 (29.7487) | -13.878 (43.7568) | -19.415 (32.6450) | -27.073 (41.9299)
  Week 8: number analyzed (Participants) | 41 | 39 | 40 | 38 | 41
  Week 8 | 1.561 (29.1042) | -12.077 (28.9876) | -5.475 (44.7718) | -17.605 (29.8442) | -26.195 (44.1719)
  Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Week 12 | -2.171 (32.0795) | -17.359 (35.4308) | -11.286 (40.7451) | -10.079 (44.8977) | -23.171 (47.2995)
  Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 40
  Week 16 | -18.833 (50.4844) | -18.263 (37.3259) | -13.952 (50.7173) | -9.895 (35.3246) | -25.425 (37.6556)
  Week 20: number analyzed (Participants) | 40 | 39 | 41 | 37 | 40
  Week 20 | -18.625 (50.3988) | -23.077 (39.6534) | -10.512 (48.0755) | -15.324 (28.8329) | -22.725 (42.2502)
  Week 24: number analyzed (Participants) | 39 | 38 | 40 | 36 | 40
  Week 24 | -19.974 (49.0196) | -14.000 (37.7760) | -4.600 (49.4025) | -10.972 (36.8375) | -22.900 (47.4092)
  Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Week 28 | -24.256 (51.8001) | -16.868 (40.6635) | -7.683 (47.8155) | -12.800 (30.7904) | -19.600 (42.3052)
  Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Week 32 | -22.410 (51.9553) | -18.590 (41.7226) | -13.575 (51.9304) | -20.618 (38.8969) | -23.179 (42.2018)
  Week 36: number analyzed (Participants) | 38 | 38 | 41 | 33 | 39
  Week 36 | -25.000 (52.6990) | -16.474 (46.8844) | -14.561 (50.2106) | -18.848 (40.0563) | -23.846 (45.1340)
  Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 38
  Week 40 | -23.432 (53.2747) | -20.895 (41.4845) | -14.927 (51.2652) | -24.088 (33.4133) | -21.789 (46.1467)
  Week 44: number analyzed (Participants) | 37 | 38 | 39 | 34 | 36
  Week 44 | -22.703 (57.8383) | -22.474 (41.0627) | -18.051 (49.1646) | -24.735 (38.4710) | -31.389 (48.5306)
  Week 48: number analyzed (Participants) | 38 | 37 | 41 | 33 | 39
  Week 48 | -27.395 (56.2963) | -23.811 (47.1150) | -24.220 (46.2458) | -22.273 (37.4243) | -28.974 (42.9960)

20. Secondary Outcome: Changes From Baseline in Biochemistry Parameters During the Study (Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma Glutamyl Transferase, Lactate Dehydrogenase)
Description: Alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, gamma glutamyl transferase, lactate dehydrogenase were measured in units per liter (U/L).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
U/L
  Alanine Aminotransferase Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Alanine Aminotransferase Week 1 | -1.366 (12.7451) | 2.526 (15.5211) | 2.628 (42.1234) | 3.122 (10.2791) | 0.700 (9.5868)
  Alanine Aminotransferase Week 2 | -1.714 (15.4624) | 2.026 (8.9428) | -1.047 (41.1223) | 4.927 (20.9623) | 1.171 (10.2978)
  Alanine Aminotransferase Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Alanine Aminotransferase Week 4 | -3.854 (15.1897) | 1.553 (16.2758) | -3.952 (38.9546) | 22.756 (139.8531) | -1.561 (10.1392)
  Alanine Aminotransferase Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Alanine Aminotransferase Week 8 | -4.707 (13.6478) | -1.385 (9.4580) | 5.465 (68.0764) | 0.795 (11.4321) | -1.659 (11.1009)
  Alanine Aminotransferase Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Alanine Aminotransferase Week 12 | -4.220 (15.1765) | 0.359 (12.2356) | -4.429 (38.1756) | 1.184 (13.0692) | -1.390 (8.1941)
  Alanine Aminotransferase Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Alanine Aminotransferase Week 16 | -2.048 (18.0026) | 2.684 (16.3229) | -4.857 (38.6211) | 0.579 (12.9273) | 0.829 (11.5432)
  Alanine Aminotransferase Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Alanine Aminotransferase Week 20 | 0.300 (39.9482) | 3.821 (13.0139) | -4.881 (39.1808) | -0.838 (11.1118) | -1.350 (10.5479)
  Alanine Aminotransferase Week 24: number analyzed (Participants) | 39 | 38 | 41 | 36 | 40
  Alanine Aminotransferase Week 24 | -1.564 (19.4974) | 2.789 (14.5475) | -5.659 (39.6652) | 1.528 (11.0259) | -3.475 (8.6202)
  Alanine Aminotransferase Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Alanine Aminotransferase Week 28 | -3.385 (17.7373) | 2.658 (12.8174) | -3.244 (43.4688) | -0.171 (8.7228) | -2.775 (10.4280)
  Alanine Aminotransferase Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Alanine Aminotransferase Week 32 | -4.487 (16.5400) | 2.385 (12.8956) | -4.150 (44.0126) | -2.176 (12.7742) | -0.821 (11.5482)
  Alanine Aminotransferase Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Alanine Aminotransferase Week 36 | 0.579 (10.5411) | 0.184 (11.8660) | -2.976 (42.9275) | -0.471 (11.2848) | -1.103 (10.6296)
  Alanine Aminotransferase Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Alanine Aminotransferase Week 40 | -0.622 (10.2506) | 0.816 (12.6680) | -2.780 (44.9719) | -3.853 (11.1059) | -1.385 (13.1061)
  Alanine Aminotransferase Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Alanine Aminotransferase Week 44 | 2.649 (19.7993) | 1.474 (13.1514) | -3.415 (43.2966) | -3.882 (12.8741) | -2.692 (10.2525)
  Alanine Aminotransferase Week 48: number analyzed (Participants) | 38 | 37 | 41 | 34 | 40
  Alanine Aminotransferase Week 48 | 2.605 (14.0646) | 2.216 (12.8542) | -4.561 (43.1926) | -3.794 (13.1628) | -0.575 (9.6181)
  Alkaline Phosphatase Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Alkaline Phosphatase Week 1 | -1.098 (6.0034) | -1.342 (8.0983) | -2.721 (7.2056) | -3.244 (4.9989) | -4.275 (7.1360)
  Alkaline Phosphatase Week 2 | -1.905 (6.7960) | -3.282 (7.8370) | -4.349 (9.5963) | -4.805 (7.8237) | -3.585 (8.8430)
  Alkaline Phosphatase Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Alkaline Phosphatase Week 4 | -1.634 (9.0630) | -1.077 (10.4236) | -3.262 (9.9144) | -1.439 (18.3508) | -4.829 (10.9268)
  Alkaline Phosphatase Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Alkaline Phosphatase Week 8 | -2.220 (8.3711) | 0.308 (12.6515) | 1.233 (37.8014) | -5.026 (10.2019) | -3.585 (9.8336)
  Alkaline Phosphatase Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Alkaline Phosphatase Week 12 | -2.463 (8.8122) | -0.462 (12.1066) | -5.952 (11.0695) | -4.947 (12.0538) | -3.146 (17.2476)
  Alkaline Phosphatase Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Alkaline Phosphatase Week 16 | -8.357 (12.7276) | -0.895 (13.1515) | -7.238 (10.7722) | -4.605 (11.6539) | -1.512 (25.7722)
  Alkaline Phosphatase Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Alkaline Phosphatase Week 20 | -10.425 (14.0510) | -5.410 (15.1895) | -10.143 (13.0264) | -7.027 (11.8544) | -6.650 (14.8143)
  Alkaline Phosphatase Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Alkaline Phosphatase Week 24 | -12.795 (15.4752) | -4.769 (13.8097) | -9.463 (11.3448) | -6.361 (12.7843) | -7.225 (18.4231)
  Alkaline Phosphatase Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Alkaline Phosphatase Week 28 | -12.795 (16.9351) | -5.684 (15.7259) | -11.244 (12.6249) | -8.314 (10.9054) | -8.525 (16.8523)
  Alkaline Phosphatase Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Alkaline Phosphatase Week 32 | -13.667 (16.1870) | -4.769 (16.1530) | -10.900 (13.0026) | -9.118 (12.5765) | -8.385 (17.5988)
  Alkaline Phosphatase Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Alkaline Phosphatase Week 36 | -11.816 (19.2436) | -6.368 (15.4735) | -11.122 (12.3495) | -8.059 (9.5217) | -6.487 (19.2434)
  Alkaline Phosphatase Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Alkaline Phosphatase Week 40 | -11.000 (16.9706) | -5.658 (15.7485) | -11.024 (12.9180) | -10.559 (11.6987) | -8.175 (17.8884)
  Alkaline Phosphatase Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Alkaline Phosphatase Week 44 | -12.622 (17.6373) | -6.421 (14.9099) | -10.537 (13.5759) | -8.647 (10.5483) | -8.950 (18.3162)
  Alkaline Phosphatase Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Alkaline Phosphatase Week 48 | -12.211 (19.0379) | -6.500 (16.5313) | -11.049 (14.4827) | -7.765 (12.3290) | -7.875 (20.1370)
  Aspartate Aminotransferase Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Aspartate Aminotransferase Week 1 | -2.854 (10.3212) | 1.447 (6.2155) | -0.023 (27.5409) | 2.244 (6.7889) | 0.475 (5.2963)
  Aspartate Aminotransferase Week 2 | -1.762 (10.5294) | 0.487 (4.0967) | -2.233 (26.3266) | 3.805 (14.7635) | 0.780 (6.1746)
  Aspartate Aminotransferase Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Aspartate Aminotransferase Week 4 | -3.976 (10.6642) | 1.289 (7.5584) | -3.262 (25.1047) | 8.927 (52.0660) | -1.195 (4.2791)
  Aspartate Aminotransferase Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Aspartate Aminotransferase Week 8 | -3.537 (10.5477) | -0.077 (5.8687) | 2.279 (34.7805) | 1.410 (5.5900) | 0.366 (6.1877)
  Aspartate Aminotransferase Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Aspartate Aminotransferase Week 12 | -3.049 (12.2106) | 0.436 (5.3054) | -2.595 (22.5324) | 1.053 (6.9006) | 1.122 (6.2897)
  Aspartate Aminotransferase Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Aspartate Aminotransferase Week 16 | -1.048 (12.1313) | 2.974 (8.3649) | -2.595 (24.3852) | 1.526 (6.6688) | 2.122 (6.1733)
  Aspartate Aminotransferase Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Aspartate Aminotransferase Week 20 | 6.375 (60.1309) | 2.821 (6.6367) | -1.095 (25.1317) | 1.324 (7.1065) | 0.500 (4.8569)
  Aspartate Aminotransferase Week 24: number analyzed (Participants) | 39 | 38 | 41 | 36 | 40
  Aspartate Aminotransferase Week 24 | 1.718 (23.7940) | 2.237 (6.9182) | -1.902 (26.1054) | 2.889 (6.2554) | 0.325 (4.3759)
  Aspartate Aminotransferase Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Aspartate Aminotransferase Week 28 | -1.179 (13.4905) | 2.289 (6.9512) | -1.805 (27.4583) | 2.229 (6.3063) | 0.175 (4.1255)
  Aspartate Aminotransferase Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Aspartate Aminotransferase Week 32 | -1.385 (12.2895) | 1.949 (6.2826) | -0.575 (28.3177) | 0.324 (6.2654) | 2.051 (4.9997)
  Aspartate Aminotransferase Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Aspartate Aminotransferase Week 36 | 0.711 (7.3113) | 1.026 (5.5140) | -1.220 (25.5798) | 1.588 (6.6017) | 1.667 (6.0755)
  Aspartate Aminotransferase Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Aspartate Aminotransferase Week 40 | 0.946 (12.1494) | 1.316 (5.5269) | 0.244 (29.2701) | -0.647 (6.0597) | 2.462 (8.4972)
  Aspartate Aminotransferase Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Aspartate Aminotransferase Week 44 | 2.838 (15.4641) | 2.553 (7.9175) | -1.268 (28.4280) | -0.588 (7.7190) | 1.590 (6.9347)
  Aspartate Aminotransferase Week 48: number analyzed (Participants) | 38 | 37 | 41 | 34 | 40
  Aspartate Aminotransferase Week 48 | 2.158 (9.7939) | 3.459 (6.3403) | -1.927 (28.3182) | 0.441 (6.6796) | 2.900 (6.2339)
  Gamma Glutamyl Transferase Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Gamma Glutamyl Transferase Week 1 | 0.171 (5.4447) | -2.737 (7.0354) | -0.535 (10.8745) | 0.171 (5.0245) | -2.300 (6.2684)
  Gamma Glutamyl Transferase Week 2 | -0.190 (5.8736) | -2.026 (7.6828) | -4.116 (25.7527) | -0.341 (5.2517) | -1.268 (7.8773)
  Gamma Glutamyl Transferase Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Gamma Glutamyl Transferase Week 4 | -0.220 (7.2129) | -2.641 (9.9167) | -6.143 (35.5504) | 1.171 (17.6265) | 0.512 (16.3968)
  Gamma Glutamyl Transferase Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Gamma Glutamyl Transferase Week 8 | -1.829 (5.9745) | -4.410 (11.6319) | 11.581 (103.8974) | -1.795 (5.7454) | -1.805 (9.0698)
  Gamma Glutamyl Transferase Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Gamma Glutamyl Transferase Week 12 | -0.585 (5.9033) | -2.154 (10.7643) | -5.762 (34.8767) | -0.447 (8.3785) | 3.244 (21.8229)
  Gamma Glutamyl Transferase Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Gamma Glutamyl Transferase Week 16 | -0.357 (9.6445) | -1.842 (13.4476) | -4.357 (34.0020) | -0.947 (8.1868) | 15.024 (77.1617)
  Gamma Glutamyl Transferase Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Gamma Glutamyl Transferase Week 20 | -0.750 (9.5051) | -2.769 (13.0555) | -5.452 (32.1970) | -1.649 (5.5137) | 1.475 (22.2722)
  Gamma Glutamyl Transferase Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Gamma Glutamyl Transferase Week 24 | -0.615 (12.4173) | -2.769 (10.9339) | -4.122 (36.6832) | -2.639 (9.4360) | -2.625 (10.3272)
  Gamma Glutamyl Transferase Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Gamma Glutamyl Transferase Week 28 | -0.462 (11.5618) | -2.132 (11.7638) | -6.341 (36.7434) | -2.629 (7.6354) | -0.200 (11.5585)
  Gamma Glutamyl Transferase Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Gamma Glutamyl Transferase Week 32 | 0.359 (15.7872) | -1.538 (13.2463) | -7.875 (36.9103) | -3.676 (8.6435) | 2.795 (21.1501)
  Gamma Glutamyl Transferase Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Gamma Glutamyl Transferase Week 36 | -0.026 (14.7162) | -4.289 (11.4559) | -8.195 (38.6899) | -2.735 (7.1236) | 1.410 (18.0200)
  Gamma Glutamyl Transferase Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Gamma Glutamyl Transferase Week 40 | -2.568 (9.3676) | -3.842 (13.9275) | -9.073 (40.5792) | -4.088 (7.5573) | 0.925 (20.1066)
  Gamma Glutamyl Transferase Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Gamma Glutamyl Transferase Week 44 | 1.081 (23.2108) | -1.289 (21.3730) | -7.488 (34.4145) | -3.824 (7.0430) | -0.949 (11.5643)
  Gamma Glutamyl Transferase Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Gamma Glutamyl Transferase Week 48 | 1.474 (17.6723) | -2.184 (12.0850) | -7.805 (35.4924) | -2.941 (8.8247) | 2.525 (20.6112)
  Lactate Dehydrogenase Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Lactate Dehydrogenase Week 1 | -7.000 (16.1509) | 0.026 (19.6118) | -1.163 (33.1669) | -0.585 (16.6673) | -1.075 (18.4341)
  Lactate Dehydrogenase Week 2 | -5.929 (18.4858) | -0.410 (14.9045) | -5.930 (32.8325) | -2.439 (19.2146) | 0.537 (19.7270)
  Lactate Dehydrogenase Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Lactate Dehydrogenase Week 4 | -5.634 (25.5693) | 4.846 (21.4372) | -6.190 (29.5265) | 0.854 (26.6238) | -4.293 (17.4732)
  Lactate Dehydrogenase Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Lactate Dehydrogenase Week 8 | -3.561 (17.3249) | 0.026 (19.0449) | 0.140 (38.8413) | 3.513 (18.6503) | 1.439 (24.0230)
  Lactate Dehydrogenase Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Lactate Dehydrogenase Week 12 | -0.927 (28.3058) | 4.077 (21.0905) | 2.119 (27.5134) | 3.342 (17.0346) | 1.049 (22.9303)
  Lactate Dehydrogenase Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Lactate Dehydrogenase Week 16 | 0.881 (26.0180) | 15.447 (62.0267) | -4.381 (35.9600) | 0.474 (19.8967) | 1.488 (21.8325)
  Lactate Dehydrogenase Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Lactate Dehydrogenase Week 20 | 1.200 (35.1817) | 2.154 (22.8825) | 2.500 (31.6145) | 0.676 (20.9206) | 2.025 (23.0401)
  Lactate Dehydrogenase Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Lactate Dehydrogenase Week 24 | 4.462 (31.9282) | 1.333 (22.1862) | 2.878 (44.9662) | 1.944 (23.5638) | 8.550 (25.3093)
  Lactate Dehydrogenase Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Lactate Dehydrogenase Week 28 | 1.436 (21.1122) | -4.763 (21.2138) | -2.902 (34.3590) | 8.143 (44.0929) | 1.250 (22.0962)
  Lactate Dehydrogenase Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Lactate Dehydrogenase Week 32 | -6.333 (23.0587) | -6.410 (23.8324) | -4.525 (35.2762) | -2.971 (27.9171) | -1.615 (24.8052)
  Lactate Dehydrogenase Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Lactate Dehydrogenase Week 36 | 0.553 (37.3889) | -4.658 (16.8383) | -7.585 (35.0442) | -6.147 (21.6895) | 5.436 (30.0436)
  Lactate Dehydrogenase Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Lactate Dehydrogenase Week 40 | -0.216 (34.5214) | -8.289 (17.4896) | -6.366 (36.6898) | -10.618 (24.4293) | 0.000 (29.3852)
  Lactate Dehydrogenase Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Lactate Dehydrogenase Week 44 | -0.757 (32.2847) | -5.316 (21.4805) | -5.000 (34.6259) | -5.059 (22.2683) | 1.675 (24.9588)
  Lactate Dehydrogenase Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Lactate Dehydrogenase Week 48 | 4.447 (34.3493) | -1.395 (23.8061) | -4.707 (38.6654) | -7.441 (23.0443) | 4.500 (37.8120)

21. Secondary Outcome: Changes From Baseline in Biochemistry Parameters During the Study (Albumin)
Description: Albumin was measured in grams per liter (g/L).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
g/L
  Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Week 1 | -1.000 (1.7464) | -0.079 (2.1357) | 0.279 (1.8038) | -0.439 (1.8715) | -0.350 (1.6259)
  Week 2 | -0.500 (2.0982) | 0.051 (1.5719) | 0.419 (1.9908) | -0.537 (2.0988) | -0.073 (1.8220)
  Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Week 4 | -0.683 (2.4743) | 0.538 (2.1007) | 0.595 (1.9514) | -0.171 (1.9862) | 0.220 (1.9687)
  Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Week 8 | -0.634 (2.0094) | 0.154 (2.1829) | 0.581 (2.0843) | 0.077 (2.2051) | 0.195 (1.7638)
  Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Week 12 | 0.073 (2.4020) | 0.538 (2.1986) | 0.857 (1.8685) | 0.211 (1.9474) | 0.415 (2.1210)
  Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Week 16 | 0.833 (1.8468) | 1.132 (2.2800) | 0.881 (2.0025) | 0.316 (2.0678) | 0.683 (1.9422)
  Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Week 20 | 0.175 (1.9333) | 0.487 (2.4047) | 0.976 (1.7873) | -0.081 (2.1000) | 0.575 (1.8659)
  Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Week 24 | 0.385 (1.7262) | 0.949 (2.3164) | 1.341 (1.8790) | 0.722 (2.2502) | 0.875 (2.3004)
  Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Week 28 | -0.462 (2.0881) | 0.632 (2.1362) | 0.976 (1.9169) | 0.114 (1.9819) | 0.525 (2.0999)
  Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Week 32 | -0.179 (1.7452) | 0.359 (1.8706) | 0.700 (1.9897) | -0.235 (1.6341) | 0.667 (1.9912)
  Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Week 36 | -0.289 (2.6397) | 0.816 (1.7220) | 0.659 (1.6064) | -0.029 (2.0815) | 0.436 (1.9166)
  Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Week 40 | -0.108 (2.0109) | 0.763 (1.9650) | 0.805 (1.8196) | 0.000 (1.8749) | 0.400 (1.9716)
  Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Week 44 | -0.297 (2.0120) | 0.132 (2.3269) | 0.659 (2.2429) | -0.206 (1.9661) | 0.175 (2.2858)
  Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Week 48 | 0.132 (2.2800) | 0.632 (2.9903) | 0.366 (3.1682) | 0.088 (2.6671) | 0.150 (2.3044)

22. Secondary Outcome: Changes From Baseline in Biochemistry Parameters During the Study (Bilirubin, Creatinine, Urate)
Description: Bilirubin, creatinine, urate were measured in micromols per liter (μmol/L).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
μmol/L
  Bilirubin Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Bilirubin Week 1 | -0.841 (2.8968) | -1.195 (3.1083) | -0.465 (3.4868) | 0.471 (3.0332) | 0.385 (2.2726)
  Bilirubin Week 2 | -0.762 (2.9415) | 0.492 (3.1202) | 0.516 (2.7030) | 0.978 (2.9538) | 1.395 (4.0672)
  Bilirubin Week 4: number analyzed (Participants) | 41 | 38 | 42 | 41 | 41
  Bilirubin Week 4 | -0.290 (3.4900) | 0.789 (2.8952) | -0.119 (3.2318) | 1.066 (3.4454) | 1.344 (3.7625)
  Bilirubin Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Bilirubin Week 8 | -0.776 (3.7242) | 0.541 (3.1822) | 0.442 (3.8005) | 0.972 (3.4557) | 0.639 (2.8243)
  Bilirubin Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Bilirubin Week 12 | -0.261 (2.6113) | 0.341 (3.0050) | 0.095 (2.5793) | 0.629 (3.2367) | 2.073 (4.0034)
  Bilirubin Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Bilirubin Week 16 | 0.607 (3.7361) | 0.637 (3.7786) | 0.740 (3.2505) | 1.092 (3.7662) | 2.024 (3.7217)
  Bilirubin Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Bilirubin Week 20 | -0.007 (3.3543) | 0.136 (3.4239) | 1.062 (3.8164) | 1.030 (3.8636) | 1.225 (2.9632)
  Bilirubin Week 24: number analyzed (Participants) | 39 | 38 | 41 | 36 | 40
  Bilirubin Week 24 | 0.146 (3.2508) | 0.592 (4.4981) | 0.383 (3.1235) | 1.081 (2.8708) | 1.128 (2.8112)
  Bilirubin Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Bilirubin Week 28 | -0.200 (3.6974) | -0.068 (3.8885) | 0.105 (2.5550) | 0.449 (3.4106) | 1.595 (3.4093)
  Bilirubin Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Bilirubin Week 32 | 0.233 (3.2668) | 0.262 (3.7358) | 0.655 (3.1125) | 0.994 (2.6879) | 1.669 (4.0868)
  Bilirubin Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Bilirubin Week 36 | 0.942 (3.6870) | 0.776 (4.3703) | 0.078 (3.8443) | 1.012 (3.5311) | 1.095 (2.3971)
  Bilirubin Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Bilirubin Week 40 | 0.600 (3.8064) | 0.679 (3.4707) | 0.415 (3.3481) | 1.065 (3.1718) | 1.433 (3.3425)
  Bilirubin Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Bilirubin Week 44 | -0.019 (3.6800) | -0.276 (3.1827) | -0.102 (3.1253) | 0.871 (2.8347) | 1.851 (3.7976)
  Bilirubin Week 48: number analyzed (Participants) | 38 | 37 | 41 | 34 | 40
  Bilirubin Week 48 | 0.716 (4.0370) | 0.559 (3.2460) | 0.285 (3.8393) | 1.124 (3.2882) | 1.160 (3.9493)
  Creatinine Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Creatinine Week 1 | -0.512 (6.6788) | 0.368 (7.3757) | 2.442 (7.8628) | 1.366 (8.9044) | 1.300 (6.7300)
  Creatinine Week 2 | 2.310 (11.1300) | 0.026 (6.1194) | 2.093 (8.4426) | 2.537 (6.8304) | 3.317 (6.7470)
  Creatinine Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Creatinine Week 4 | 0.854 (10.2508) | 1.256 (7.0812) | 1.762 (8.8229) | -0.561 (7.3418) | 2.171 (6.9279)
  Creatinine Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Creatinine Week 8 | 1.366 (8.3269) | 1.487 (8.3756) | 3.674 (10.1997) | 1.590 (7.9131) | 3.073 (5.7810)
  Creatinine Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Creatinine Week 12 | 1.268 (8.0282) | 0.949 (8.6113) | 6.214 (9.5062) | 1.947 (9.1236) | 2.220 (8.2417)
  Creatinine Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Creatinine Week 16 | 1.833 (8.4678) | 1.421 (10.7945) | 3.738 (7.7964) | 0.658 (8.7897) | 3.976 (8.2719)
  Creatinine Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Creatinine Week 20 | 3.150 (8.3468) | 1.051 (7.7966) | 4.976 (10.5818) | 2.270 (8.5461) | 4.525 (7.4144)
  Creatinine Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Creatinine Week 24 | 1.359 (8.1741) | 0.103 (6.8817) | 3.829 (11.4256) | 1.972 (9.3914) | 4.650 (7.2627)
  Creatinine Week 28: number analyzed (Participants) | 38 | 38 | 41 | 35 | 40
  Creatinine Week 28 | 2.921 (7.0227) | 1.737 (7.4858) | 4.634 (8.9576) | 1.371 (8.3634) | 4.900 (7.2388)
  Creatinine Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Creatinine Week 32 | 1.718 (8.8227) | 2.462 (9.1360) | 2.500 (8.9299) | 4.118 (12.0825) | 4.974 (7.7408)
  Creatinine Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Creatinine Week 36 | 0.289 (7.5656) | 1.632 (7.1600) | 1.024 (8.8218) | 1.853 (10.8492) | 3.462 (6.8127)
  Creatinine Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Creatinine Week 40 | 3.838 (9.5205) | 2.974 (7.3796) | 4.122 (9.7575) | 0.647 (10.7672) | 3.200 (7.0208)
  Creatinine Week 44: number analyzed (Participants) | 35 | 36 | 41 | 33 | 40
  Creatinine Week 44 | 4.543 (10.6670) | 4.250 (8.7876) | 3.659 (8.5311) | 3.364 (10.6853) | 3.925 (8.0012)
  Creatinine Week 48: number analyzed (Participants) | 35 | 33 | 39 | 33 | 39
  Creatinine Week 48 | 3.000 (10.3299) | 4.667 (8.5355) | 3.923 (7.7371) | 2.879 (9.8513) | 3.256 (7.0290)
  Urate Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Urate Week 1 | -1.220 (37.4503) | -0.237 (43.0100) | 11.953 (60.5652) | 8.732 (39.4088) | 11.650 (61.0924)
  Urate Week 2 | 12.405 (47.5795) | -2.974 (44.8826) | 9.791 (61.4009) | 9.073 (39.3430) | 15.610 (49.0693)
  Urate Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Urate Week 4 | 10.171 (41.5493) | 0.308 (47.3193) | 13.452 (49.1633) | 5.659 (31.2591) | -4.293 (47.5753)
  Urate Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Urate Week 8 | 5.415 (42.9500) | -6.231 (40.4198) | 11.791 (64.9910) | 3.410 (33.9518) | 8.024 (44.0043)
  Urate Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Urate Week 12 | 10.707 (40.2208) | 6.795 (54.4814) | 13.881 (55.3332) | 7.553 (33.4904) | 2.805 (37.6651)
  Urate Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Urate Week 16 | 25.810 (44.1965) | 8.079 (50.0062) | 15.357 (59.0311) | 14.026 (40.5173) | 21.683 (41.1670)
  Urate Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Urate Week 20 | 28.950 (53.8602) | 4.692 (59.0420) | 16.048 (63.4346) | 10.622 (42.1567) | 10.600 (44.3262)
  Urate Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Urate Week 24 | 17.410 (45.0045) | 9.923 (54.9648) | 3.683 (58.6977) | 6.667 (45.2580) | 6.950 (45.8638)
  Urate Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Urate Week 28 | -0.897 (29.4331) | 9.447 (59.8655) | 18.976 (62.4894) | -6.371 (40.1227) | 1.250 (45.8972)
  Urate Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Urate Week 32 | 17.026 (47.8185) | 2.821 (48.9042) | 5.800 (56.2017) | 3.971 (45.1103) | 17.077 (40.3089)
  Urate Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Urate Week 36 | 0.211 (37.5630) | -4.868 (49.1419) | -10.927 (59.4228) | 4.735 (42.4309) | 5.846 (49.4259)
  Urate Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Urate Week 40 | 9.730 (43.5295) | 15.605 (53.8931) | 9.976 (62.8739) | -5.029 (41.2630) | 7.255 (46.0833)
  Urate Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Urate Week 44 | 20.541 (57.9164) | 7.605 (64.3342) | -8.854 (67.3523) | 1.382 (47.9558) | 10.675 (50.8963)
  Urate Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Urate Week 48 | 8.684 (53.6208) | 3.895 (48.5831) | -3.220 (64.9282) | 1.853 (54.8762) | 8.050 (49.1956)

23. Secondary Outcome: Changes From Baseline in Biochemistry Parameters During the Study (Calcium, Chloride, Cholesterol, Glucose, Magnesium, Potassium, Sodium)
Description: Calcium, chloride, cholesterol, glucose, magnesium, potassium, sodium were measured in millimoles per liter (mmol/L).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
mmol/L
  Calcium Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Calcium Week 1 | -0.034 (0.0810) | -0.017 (0.0984) | -0.008 (0.0858) | -0.002 (0.0990) | -0.014 (0.0897)
  Calcium Week 2 | -0.021 (0.0951) | 0.002 (0.0973) | 0.009 (0.1304) | -0.024 (0.1001) | -0.022 (0.0938)
  Calcium Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Calcium Week 4 | -0.029 (0.1079) | -0.011 (0.1015) | -0.021 (0.0973) | -0.047 (0.1147) | -0.020 (0.0917)
  Calcium Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Calcium Week 8 | -0.024 (0.0942) | -0.006 (0.0926) | 0.008 (0.1260) | -0.004 (0.1105) | -0.022 (0.0975)
  Calcium Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Calcium Week 12 | -0.021 (0.1009) | -0.025 (0.1090) | 0.021 (0.1057) | -0.020 (0.1088) | -0.025 (0.0923)
  Calcium Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Calcium Week 16 | 0.004 (0.0826) | -0.006 (0.1079) | 0.023 (0.1334) | -0.004 (0.1027) | 0.005 (0.0888)
  Calcium Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Calcium Week 20 | 0.002 (0.0931) | 0.000 (0.1013) | 0.017 (0.0999) | -0.008 (0.0948) | -0.018 (0.0919)
  Calcium Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Calcium Week 24 | 0.011 (0.1019) | -0.002 (0.1028) | 0.015 (0.0845) | 0.004 (0.0896) | 0.003 (0.0974)
  Calcium Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Calcium Week 28 | -0.027 (0.1117) | 0.002 (0.0877) | 0.009 (0.1068) | 0.008 (0.0909) | -0.021 (0.1043)
  Calcium Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Calcium Week 32 | -0.023 (0.1069) | 0.000 (0.0952) | 0.001 (0.1074) | -0.017 (0.0932) | -0.008 (0.1024)
  Calcium Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Calcium Week 36 | -0.013 (0.1172) | 0.007 (0.0804) | -0.005 (0.1096) | 0.001 (0.0972) | -0.015 (0.0936)
  Calcium Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Calcium Week 40 | 0.003 (0.0905) | 0.001 (0.0807) | -0.007 (0.1084) | -0.019 (0.0809) | -0.025 (0.0947)
  Calcium Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Calcium Week 44 | -0.027 (0.0920) | -0.018 (0.0861) | -0.008 (0.1023) | -0.019 (0.0839) | -0.042 (0.0972)
  Calcium Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Calcium Week 48 | -0.010 (0.0881) | -0.009 (0.1033) | -0.014 (0.1126) | -0.014 (0.0912) | -0.034 (0.0861)
  Chloride Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Chloride Week 1 | -0.195 (2.1121) | -0.105 (2.5446) | -0.674 (4.1388) | -0.244 (2.5572) | -0.125 (2.3986)
  Chloride Week 2 | -0.214 (2.1131) | 0.308 (2.6273) | 0.093 (2.7500) | 0.415 (2.5296) | -0.439 (2.4192)
  Chloride Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Chloride Week 4 | -0.293 (1.9525) | -0.333 (2.2750) | 0.000 (2.4792) | 0.024 (2.6409) | 0.000 (2.6363)
  Chloride Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Chloride Week 8 | -0.537 (2.1920) | 0.615 (2.4346) | 0.047 (2.6988) | 0.538 (2.3038) | 0.683 (2.4025)
  Chloride Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Chloride Week 12 | 0.341 (2.2205) | -0.282 (2.3946) | 0.548 (2.5681) | -0.211 (2.3499) | 0.000 (2.4393)
  Chloride Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Chloride Week 16 | -0.310 (1.8934) | 0.026 (2.2837) | 0.190 (2.0864) | -0.184 (2.2644) | -0.268 (2.1334)
  Chloride Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Chloride Week 20 | -0.325 (2.4640) | -0.538 (2.1502) | 0.262 (2.3484) | 0.162 (2.6616) | 0.075 (2.3685)
  Chloride Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Chloride Week 24 | -0.615 (2.0081) | -0.128 (2.5462) | -0.390 (2.6351) | -0.306 (2.1885) | -0.050 (2.5415)
  Chloride Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Chloride Week 28 | 0.128 (2.3190) | 0.000 (2.6913) | 0.195 (2.3154) | 0.086 (2.5365) | 0.250 (2.5090)
  Chloride Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Chloride Week 32 | -0.154 (2.2069) | 0.436 (2.3708) | 0.500 (2.2072) | 0.794 (2.3196) | 0.282 (2.0641)
  Chloride Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Chloride Week 36 | 0.237 (1.9923) | 0.684 (2.4285) | 0.732 (1.9239) | 0.294 (2.5999) | 0.205 (2.4299)
  Chloride Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Chloride Week 40 | -0.054 (2.5380) | 0.263 (2.6271) | 0.707 (2.4418) | 0.824 (2.4676) | 0.500 (2.4495)
  Chloride Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Chloride Week 44 | 0.135 (1.9027) | 0.579 (2.6977) | 0.756 (2.1069) | 0.882 (2.8044) | 0.200 (2.5840)
  Chloride Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Chloride Week 48 | 0.605 (2.0994) | 0.737 (2.8158) | 1.024 (2.4545) | 0.971 (2.5044) | 0.725 (2.7826)
  Cholesterol Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Cholesterol Week 1 | -0.254 (0.4371) | 0.032 (0.4307) | 0.244 (0.5220) | 0.105 (0.4690) | 0.102 (0.3965)
  Cholesterol Week 2 | -0.224 (0.4154) | 0.108 (0.5132) | 0.295 (0.5178) | 0.054 (0.5441) | 0.222 (0.6101)
  Cholesterol Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Cholesterol Week 4 | -0.198 (0.6334) | -0.023 (0.5905) | 0.210 (0.8027) | 0.093 (0.6525) | 0.151 (0.4178)
  Cholesterol Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Cholesterol Week 8 | -0.190 (0.6935) | -0.023 (0.5770) | 0.284 (0.8012) | 0.074 (0.7920) | 0.061 (0.6268)
  Cholesterol Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Cholesterol Week 12 | -0.124 (0.6719) | 0.013 (0.7473) | 0.117 (0.7616) | 0.005 (0.6045) | 0.212 (0.7491)
  Cholesterol Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Cholesterol Week 16 | 0.095 (0.6811) | 0.184 (0.6378) | 0.138 (0.6814) | 0.068 (0.6014) | 0.249 (0.7075)
  Cholesterol Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Cholesterol Week 20 | 0.053 (0.7609) | 0.126 (0.6889) | 0.186 (0.9669) | 0.116 (0.7101) | 0.115 (0.7718)
  Cholesterol Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Cholesterol Week 24 | 0.041 (0.8729) | 0.013 (0.8673) | 0.127 (1.0682) | -0.003 (0.6984) | 0.077 (0.5686)
  Cholesterol Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Cholesterol Week 28 | -0.044 (0.9797) | -0.037 (0.8930) | 0.076 (1.1434) | -0.037 (0.5801) | 0.100 (0.5923)
  Cholesterol Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Cholesterol Week 32 | -0.085 (0.8540) | -0.079 (0.8918) | 0.175 (1.0895) | -0.050 (0.5945) | 0.256 (0.6920)
  Cholesterol Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Cholesterol Week 36 | 0.005 (0.7322) | 0.024 (0.7951) | 0.117 (0.8408) | -0.038 (0.6597) | 0.144 (0.7950)
  Cholesterol Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Cholesterol Week 40 | -0.103 (0.7541) | -0.118 (0.9109) | 0.183 (0.8947) | -0.135 (0.7454) | 0.110 (0.7824)
  Cholesterol Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Cholesterol Week 44 | -0.170 (0.8082) | -0.176 (1.0874) | 0.071 (0.9341) | -0.218 (0.9150) | -0.000 (0.8407)
  Cholesterol Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Cholesterol Week 48 | -0.282 (0.7891) | -0.279 (0.8348) | 0.012 (0.8883) | -0.253 (0.6653) | -0.083 (0.5817)
  Glucose Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Glucose Week 1 | 0.307 (1.3942) | 0.103 (0.7027) | 0.077 (1.1366) | 0.173 (1.0232) | -0.060 (0.8445)
  Glucose Week 2 | 0.062 (0.6681) | 0.013 (0.8348) | 0.221 (0.9652) | 0.129 (1.2364) | 0.190 (0.8938)
  Glucose Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Glucose Week 4 | 0.298 (0.8575) | 0.015 (0.6888) | 0.248 (0.7693) | 0.249 (1.0659) | 0.134 (0.7428)
  Glucose Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Glucose Week 8 | 0.112 (0.9127) | 0.308 (0.7696) | 0.258 (0.9254) | 0.344 (0.6939) | 0.256 (0.7075)
  Glucose Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Glucose Week 12 | 0.110 (0.9146) | 0.005 (0.6117) | 0.188 (0.7533) | 0.111 (0.6455) | -0.124 (0.6636)
  Glucose Week 16: number analyzed (Participants) | 42 | 37 | 42 | 38 | 41
  Glucose Week 16 | 0.176 (0.8363) | 0.195 (0.6316) | 0.424 (1.1521) | 0.276 (0.8280) | 0.398 (0.8332)
  Glucose Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Glucose Week 20 | 0.208 (1.0560) | 0.315 (1.0225) | 0.267 (1.0132) | 0.632 (0.9741) | 0.165 (1.0366)
  Glucose Week 24: number analyzed (Participants) | 39 | 39 | 40 | 36 | 40
  Glucose Week 24 | 0.018 (1.1856) | 0.092 (0.7747) | 0.328 (0.8554) | 0.061 (1.0462) | 0.037 (0.6295)
  Glucose Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Glucose Week 28 | 0.246 (1.1812) | 0.263 (0.9371) | 0.322 (1.1372) | 0.263 (1.0053) | 0.262 (0.6412)
  Glucose Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Glucose Week 32 | 0.333 (1.2671) | 0.236 (0.7013) | 0.570 (1.0301) | 0.356 (1.1021) | 0.203 (0.5945)
  Glucose Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Glucose Week 36 | 0.089 (0.9061) | 0.342 (0.9406) | 0.234 (1.0379) | 0.174 (1.0175) | 0.290 (0.7789)
  Glucose Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Glucose Week 40 | 0.143 (1.0885) | 0.245 (1.1081) | 0.507 (1.1257) | 0.203 (0.7420) | 0.125 (0.7016)
  Glucose Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Glucose Week 44 | 0.222 (1.4919) | 0.200 (1.0950) | 0.185 (0.8688) | 0.303 (1.2760) | 0.197 (0.8966)
  Glucose Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Glucose Week 48 | -0.013 (1.2512) | 0.045 (0.8472) | 0.141 (0.9341) | 0.276 (1.0841) | 0.100 (0.7835)
  Magnesium Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Magnesium Week 1 | -0.010 (0.0672) | -0.007 (0.0676) | 0.002 (0.0694) | -0.014 (0.0573) | -0.015 (0.0680)
  Magnesium Week 2 | -0.004 (0.0795) | 0.008 (0.0745) | -0.011 (0.0771) | -0.019 (0.0624) | -0.007 (0.0680)
  Magnesium Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Magnesium Week 4 | -0.022 (0.0606) | 0.009 (0.0725) | -0.012 (0.0789) | -0.020 (0.0712) | -0.005 (0.0998)
  Magnesium Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Magnesium Week 8 | -0.016 (0.0706) | -0.008 (0.0593) | -0.013 (0.0819) | -0.015 (0.0706) | -0.006 (0.0624)
  Magnesium Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Magnesium Week 12 | 0.010 (0.0797) | 0.008 (0.0847) | -0.011 (0.0733) | -0.001 (0.0660) | 0.003 (0.0730)
  Magnesium Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Magnesium Week 16 | -0.002 (0.0742) | 0.003 (0.0823) | -0.021 (0.0659) | -0.009 (0.0629) | -0.002 (0.0731)
  Magnesium Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Magnesium Week 20 | -0.007 (0.0811) | -0.012 (0.0728) | -0.018 (0.0659) | -0.005 (0.0724) | -0.009 (0.0636)
  Magnesium Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Magnesium Week 24 | -0.005 (0.0757) | -0.004 (0.0572) | -0.014 (0.0732) | -0.009 (0.0559) | -0.016 (0.0664)
  Magnesium Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Magnesium Week 28 | -0.027 (0.0713) | -0.007 (0.0525) | -0.018 (0.0678) | -0.019 (0.0719) | -0.017 (0.0565)
  Magnesium Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Magnesium Week 32 | -0.023 (0.0727) | -0.016 (0.0641) | -0.016 (0.0603) | -0.012 (0.0670) | -0.013 (0.0572)
  Magnesium Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Magnesium Week 36 | -0.015 (0.0694) | -0.001 (0.0596) | -0.031 (0.0698) | -0.004 (0.0534) | -0.007 (0.0563)
  Magnesium Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Magnesium Week 40 | -0.032 (0.0681) | -0.007 (0.0541) | -0.014 (0.0754) | -0.024 (0.0636) | -0.009 (0.0684)
  Magnesium Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Magnesium Week 44 | -0.024 (0.0677) | -0.000 (0.0597) | -0.009 (0.0685) | -0.024 (0.0668) | -0.016 (0.0667)
  Magnesium Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Magnesium Week 48 | -0.004 (0.0633) | -0.004 (0.0546) | -0.014 (0.0569) | -0.006 (0.0616) | -0.009 (0.0648)
  Potassium Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Potassium Week 1 | -0.095 (0.2701) | 0.089 (0.3608) | 0.081 (0.4289) | -0.017 (0.3098) | -0.062 (0.3216)
  Potassium Week 2 | -0.098 (0.2975) | 0.085 (0.4095) | 0.002 (0.3327) | -0.005 (0.3521) | 0.027 (0.3074)
  Potassium Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Potassium Week 4 | -0.080 (0.2522) | 0.008 (0.3821) | 0.026 (0.2632) | 0.024 (0.4030) | -0.063 (0.2853)
  Potassium Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Potassium Week 8 | -0.056 (0.2907) | 0.069 (0.3221) | 0.014 (0.3306) | -0.010 (0.3135) | 0.000 (0.2520)
  Potassium Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Potassium Week 12 | -0.073 (0.3217) | 0.033 (0.3398) | -0.024 (0.3192) | -0.082 (0.3074) | -0.080 (0.2977)
  Potassium Week 16: number analyzed (Participants) | 42 | 36 | 42 | 38 | 41
  Potassium Week 16 | -0.086 (0.3258) | 0.083 (0.3112) | 0.012 (0.3651) | -0.037 (0.3035) | -0.020 (0.2713)
  Potassium Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Potassium Week 20 | -0.092 (0.3846) | 0.031 (0.3381) | 0.055 (0.3494) | -0.019 (0.3627) | 0.000 (0.2774)
  Potassium Week 24: number analyzed (Participants) | 39 | 39 | 40 | 36 | 40
  Potassium Week 24 | -0.095 (0.3308) | -0.072 (0.3052) | 0.030 (0.3844) | -0.094 (0.3414) | -0.062 (0.2967)
  Potassium Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Potassium Week 28 | -0.077 (0.3141) | 0.105 (0.3616) | 0.063 (0.4265) | -0.003 (0.3312) | -0.030 (0.3480)
  Potassium Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Potassium Week 32 | -0.062 (0.3306) | 0.069 (0.3621) | 0.023 (0.4154) | 0.056 (0.2688) | 0.046 (0.3094)
  Potassium Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Potassium Week 36 | -0.092 (0.3388) | 0.045 (0.3689) | 0.066 (0.4316) | 0.003 (0.3205) | 0.033 (0.3359)
  Potassium Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Potassium Week 40 | -0.092 (0.3616) | 0.089 (0.3826) | 0.024 (0.3484) | -0.003 (0.3407) | -0.017 (0.3456)
  Potassium Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Potassium Week 44 | -0.119 (0.2933) | 0.029 (0.3571) | 0.068 (0.4344) | 0.094 (0.3084) | -0.035 (0.3009)
  Potassium Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Potassium Week 48 | -0.137 (0.3627) | -0.053 (0.3244) | -0.032 (0.3274) | 0.003 (0.4123) | -0.027 (0.3250)
  Sodium Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Sodium Week 1 | -0.146 (1.5582) | -0.184 (1.7531) | 0.000 (2.0471) | -0.610 (2.0722) | -0.375 (2.1326)
  Sodium Week 2 | -0.500 (1.6417) | -0.513 (1.8191) | -0.209 (1.9341) | -0.244 (2.0221) | -0.341 (2.1167)
  Sodium Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Sodium Week 4 | -0.732 (1.8442) | -0.385 (1.6482) | -0.214 (2.3430) | -0.707 (2.0155) | -0.805 (1.8196)
  Sodium Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Sodium Week 8 | -0.854 (2.0070) | -0.410 (1.3711) | -0.860 (2.2316) | -0.359 (1.7394) | -0.463 (2.2924)
  Sodium Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Sodium Week 12 | -0.512 (1.8858) | -0.513 (1.4845) | -0.619 (2.0357) | -0.632 (2.1738) | -0.854 (2.3512)
  Sodium Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Sodium Week 16 | -0.738 (1.8086) | -0.211 (1.7423) | -0.714 (1.7708) | -0.842 (2.3656) | -0.780 (1.7250)
  Sodium Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Sodium Week 20 | -0.675 (1.7155) | -0.538 (1.4482) | -0.857 (2.1928) | -0.595 (2.1661) | -0.775 (1.9147)
  Sodium Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Sodium Week 24 | -0.821 (1.7751) | -0.487 (1.5196) | -0.463 (2.0137) | -0.472 (1.8124) | -0.725 (1.7393)
  Sodium Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Sodium Week 28 | -0.462 (2.2924) | -0.658 (1.8494) | -0.683 (1.8767) | -0.457 (2.3307) | -0.575 (2.5609)
  Sodium Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Sodium Week 32 | -1.077 (1.8692) | -0.128 (1.9219) | -0.525 (1.8809) | -0.441 (1.6732) | -0.667 (1.8257)
  Sodium Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Sodium Week 36 | -0.711 (2.0122) | -0.263 (1.8986) | -0.512 (1.8725) | -0.618 (1.9850) | -0.436 (2.2337)
  Sodium Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Sodium Week 40 | -0.432 (2.1153) | -0.474 (1.6397) | -0.512 (2.1578) | -0.882 (1.9812) | -0.950 (2.0248)
  Sodium Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Sodium Week 44 | -0.486 (1.8352) | -0.737 (2.0492) | -0.878 (1.9390) | -0.647 (1.8238) | -1.000 (2.4179)
  Sodium Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Sodium Week 48 | -0.237 (1.7772) | -0.763 (1.8074) | -0.732 (1.8845) | -0.706 (1.5281) | -0.750 (2.1334)

24. Secondary Outcome: Changes From Baseline in Biochemistry Parameters During the Study (Urea Nitrogen)
Description: Urea nitrogen was measured in millimoles per liter (mmol/L).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
mmol/L
  Week 1: number analyzed (Participants) | 41 | 38 | 43 | 41 | 40
  Week 1 | -0.093 (1.0815) | 0.126 (1.2116) | -0.123 (1.0989) | -0.012 (1.0900) | 0.173 (1.5513)
  Week 2 | 0.386 (1.8183) | -0.208 (1.1329) | -0.047 (1.0359) | 0.024 (1.1762) | 0.212 (1.3064)
  Week 4: number analyzed (Participants) | 41 | 39 | 42 | 41 | 41
  Week 4 | 0.027 (1.3217) | 0.013 (1.1307) | 0.083 (1.1244) | -0.224 (1.1449) | 0.007 (1.2384)
  Week 8: number analyzed (Participants) | 41 | 39 | 43 | 39 | 41
  Week 8 | 0.007 (0.9936) | 0.023 (1.1685) | -0.070 (1.1143) | -0.379 (1.2316) | 0.080 (1.1265)
  Week 12: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Week 12 | -0.166 (1.2654) | -0.244 (1.1740) | -0.231 (1.3357) | -0.429 (1.1733) | -0.151 (1.2426)
  Week 16: number analyzed (Participants) | 42 | 38 | 42 | 38 | 41
  Week 16 | -0.133 (1.0656) | -0.087 (0.9793) | -0.200 (1.3083) | -0.218 (1.0747) | 0.012 (1.1996)
  Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Week 20 | -0.207 (1.2670) | -0.490 (1.0901) | -0.064 (1.2916) | -0.357 (1.1572) | -0.035 (1.3202)
  Week 24: number analyzed (Participants) | 39 | 39 | 41 | 36 | 40
  Week 24 | -0.256 (1.1378) | -0.523 (1.1235) | -0.232 (1.4951) | -0.289 (1.1369) | -0.138 (1.2245)
  Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Week 28 | -0.267 (1.3487) | -0.287 (1.0992) | 0.012 (1.3020) | -0.263 (1.1835) | -0.082 (1.3239)
  Week 32: number analyzed (Participants) | 39 | 39 | 40 | 34 | 39
  Week 32 | -0.097 (1.0396) | -0.141 (1.3098) | -0.200 (1.1266) | -0.326 (1.1199) | 0.082 (1.1841)
  Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Week 36 | -0.203 (1.0579) | -0.308 (1.1757) | 0.015 (1.1094) | -0.247 (1.1683) | -0.018 (1.1014)
  Week 40: number analyzed (Participants) | 37 | 38 | 41 | 34 | 40
  Week 40 | -0.214 (1.2537) | 0.192 (1.3690) | 0.068 (1.1230) | -0.132 (1.1834) | 0.283 (1.3435)
  Week 44: number analyzed (Participants) | 37 | 38 | 41 | 34 | 39
  Week 44 | -0.105 (1.3389) | -0.047 (1.3456) | -0.054 (1.1276) | -0.229 (1.1979) | 0.210 (1.2264)
  Week 48: number analyzed (Participants) | 38 | 38 | 41 | 34 | 40
  Week 48 | -0.111 (1.4431) | -0.113 (1.1796) | -0.222 (1.4085) | -0.285 (1.2611) | 0.088 (1.4580)

25. Secondary Outcome: Changes From Baseline in Urinalysis Parameters During the Study (Erythrocytes, Leukocytes, Renal Epithelial Casts, Squamous Epithelial Cells, Transitional Epithelial Cells)
Description: Erythrocytes, leukocytes, renal epithelial casts, squamous epithelial cells, transitional epithelial cells were measured in cells per high power field (cells/HPF).
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP. Number of participants reflect those with non-missing urinalysis results during the study.
Measure: Mean (Standard Deviation); unit: cells/HPF
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 2 | 6 | 5 | 7 | 4
cells/HPF
  Erythrocytes Week 1: number analyzed (Participants) | 1 | 4 | 3 | 5 | 3
  Erythrocytes Week 1 | -55.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.750 (0.9574) | 0.333 (0.5774) | 0.000 (0.0000) | 0.333 (0.5774)
  Erythrocytes Week 2: number analyzed (Participants) | 1 | 4 | 4 | 4 | 3
  Erythrocytes Week 2 | -54.000 (NA) — Value was not evaluable because only one participant was analyzed. | -0.500 (0.5774) | 0.250 (0.5000) | 0.000 (0.0000) | 1.333 (2.5166)
  Erythrocytes Week 4: number analyzed (Participants) | 1 | 3 | 5 | 4 | 2
  Erythrocytes Week 4 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 3.333 (5.7735) | 0.000 (0.7071) | 0.250 (0.5000) | -0.500 (0.7071)
  Erythrocytes Week 8: number analyzed (Participants) | 0 | 3 | 4 | 2 | 3
  Erythrocytes Week 8 |  | 0.000 (0.0000) | 0.000 (0.8165) | 0.000 (0.0000) | 0.000 (1.0000)
  Erythrocytes Week 12: number analyzed (Participants) | 1 | 3 | 5 | 2 | 3
  Erythrocytes Week 12 | -23.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.800 (1.3038) | 0.000 (0.0000) | -0.333 (0.5774)
  Erythrocytes Week 16: number analyzed (Participants) | 1 | 5 | 4 | 5 | 2
  Erythrocytes Week 16 | -55.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.800 (1.7889) | 0.500 (1.7321) | 0.000 (0.0000) | 2.500 (3.5355)
  Erythrocytes Week 20: number analyzed (Participants) | 2 | 4 | 5 | 6 | 4
  Erythrocytes Week 20 | -30.000 (35.3553) | 0.000 (0.0000) | 0.400 (1.1402) | 0.000 (0.0000) | 0.250 (0.5000)
  Erythrocytes Week 24: number analyzed (Participants) | 0 | 4 | 4 | 7 | 3
  Erythrocytes Week 24 |  | -0.250 (0.5000) | 0.250 (0.5000) | -0.143 (0.8997) | 1.000 (2.6458)
  Erythrocytes Week 28: number analyzed (Participants) | 1 | 4 | 5 | 4 | 3
  Erythrocytes Week 28 | -5.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.8165) | 0.400 (1.5166) | 0.000 (0.0000) | 2.333 (5.7735)
  Erythrocytes Week 32: number analyzed (Participants) | 2 | 3 | 4 | 6 | 3
  Erythrocytes Week 32 | -27.500 (38.8909) | 0.000 (0.0000) | 0.250 (0.5000) | 0.000 (0.0000) | 2.000 (3.4641)
  Erythrocytes Week 36: number analyzed (Participants) | 1 | 6 | 4 | 1 | 1
  Erythrocytes Week 36 | -55.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.250 (0.5000) | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | -1.000 (NA) — Value was not evaluable because only one participant was analyzed.
  Erythrocytes Week 40: number analyzed (Participants) | 0 | 4 | 4 | 4 | 2
  Erythrocytes Week 40 |  | -0.250 (0.5000) | 0.750 (1.5000) | -0.250 (0.5000) | 0.000 (0.0000)
  Erythrocytes Week 44: number analyzed (Participants) | 1 | 5 | 5 | 4 | 2
  Erythrocytes Week 44 | -55.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.400 (0.8944) | -0.250 (1.2583) | 0.000 (0.0000)
  Erythrocytes Week 48: number analyzed (Participants) | 2 | 6 | 4 | 3 | 4
  Erythrocytes Week 48 | -27.500 (38.8909) | 0.167 (0.4082) | 1.750 (3.5000) | 0.000 (0.0000) | 0.000 (0.8165)
  Leukocytes Week 1: number analyzed (Participants) | 1 | 4 | 3 | 5 | 3
  Leukocytes Week 1 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 2.750 (6.1847) | -7.667 (13.2791) | -0.200 (1.0954) | 0.667 (1.1547)
  Leukocytes Week 2: number analyzed (Participants) | 1 | 4 | 4 | 4 | 3
  Leukocytes Week 2 | 2.000 (NA) — Value was not evaluable because only one participant was analyzed. | -2.500 (2.0817) | -3.000 (6.6833) | -0.250 (0.5000) | 0.000 (0.0000)
  Leukocytes Week 4: number analyzed (Participants) | 1 | 3 | 5 | 4 | 2
  Leukocytes Week 4 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | -4.600 (10.2372) | 0.250 (0.5000) | 2.000 (2.8284)
  Leukocytes Week 8: number analyzed (Participants) | 0 | 2 | 4 | 2 | 3
  Leukocytes Week 8 |  | 0.000 (0.0000) | -1.500 (3.6968) | 0.000 (0.0000) | 4.000 (6.9282)
  Leukocytes Week 12: number analyzed (Participants) | 1 | 3 | 4 | 2 | 3
  Leukocytes Week 12 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 1.667 (4.7258) | 13.500 (26.3376) | 0.000 (0.0000) | 0.000 (0.0000)
  Leukocytes Week 16: number analyzed (Participants) | 1 | 5 | 4 | 5 | 2
  Leukocytes Week 16 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | -0.200 (1.7889) | 33.750 (67.5000) | -0.400 (0.8944) | 0.500 (0.7071)
  Leukocytes Week 20: number analyzed (Participants) | 2 | 4 | 5 | 6 | 4
  Leukocytes Week 20 | 0.000 (2.8284) | 3.000 (6.0000) | 57.800 (145.4036) | 0.667 (1.5055) | -6.750 (14.8633)
  Leukocytes Week 24: number analyzed (Participants) | 0 | 4 | 4 | 7 | 3
  Leukocytes Week 24 |  | 2.750 (4.8563) | -6.500 (13.0000) | 2.286 (4.8206) | 0.333 (0.5774)
  Leukocytes Week 28: number analyzed (Participants) | 1 | 4 | 5 | 4 | 3
  Leukocytes Week 28 | -2.000 (NA) — Value was not evaluable because only one participant was analyzed. | -0.750 (0.9574) | -5.400 (12.0748) | 0.000 (0.0000) | 2.333 (4.0415)
  Leukocytes Week 32: number analyzed (Participants) | 2 | 3 | 4 | 6 | 3
  Leukocytes Week 32 | 0.000 (0.0000) | 3.333 (5.7735) | -6.500 (13.0000) | -1.333 (1.6330) | 1.333 (2.3094)
  Leukocytes Week 36: number analyzed (Participants) | 1 | 6 | 4 | 1 | 1
  Leukocytes Week 36 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.667 (2.7325) | 0.000 (0.0000) | 24.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (NA) — Value was not evaluable because only one participant was analyzed.
  Leukocytes Week 40: number analyzed (Participants) | 0 | 4 | 4 | 4 | 2
  Leukocytes Week 40 |  | -0.500 (2.5166) | -7.500 (15.0000) | 1.500 (3.0000) | 0.000 (0.0000)
  Leukocytes Week 44: number analyzed (Participants) | 1 | 5 | 5 | 4 | 2
  Leukocytes Week 44 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.400 (0.8944) | -1.400 (3.1305) | -0.500 (1.0000) | 0.000 (0.0000)
  Leukocytes Week 48: number analyzed (Participants) | 2 | 6 | 4 | 3 | 4
  Leukocytes Week 48 | 0.000 (0.0000) | 8.000 (21.6148) | 69.500 (139.0000) | -1.000 (1.7321) | 0.250 (0.5000)
  Renal Epithelial Casts Week 1: number analyzed (Participants) | 1 | 4 | 3 | 5 | 3
  Renal Epithelial Casts Week 1 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 2: number analyzed (Participants) | 1 | 4 | 4 | 4 | 3
  Renal Epithelial Casts Week 2 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 4: number analyzed (Participants) | 1 | 3 | 5 | 4 | 2
  Renal Epithelial Casts Week 4 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 8: number analyzed (Participants) | 0 | 3 | 4 | 2 | 3
  Renal Epithelial Casts Week 8 |  | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 12: number analyzed (Participants) | 1 | 3 | 5 | 2 | 3
  Renal Epithelial Casts Week 12 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 16: number analyzed (Participants) | 1 | 5 | 4 | 5 | 2
  Renal Epithelial Casts Week 16 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 20: number analyzed (Participants) | 2 | 4 | 5 | 6 | 4
  Renal Epithelial Casts Week 20 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 24: number analyzed (Participants) | 0 | 4 | 4 | 7 | 3
  Renal Epithelial Casts Week 24 |  | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 28: number analyzed (Participants) | 1 | 4 | 5 | 4 | 3
  Renal Epithelial Casts Week 28 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 32: number analyzed (Participants) | 2 | 3 | 4 | 6 | 3
  Renal Epithelial Casts Week 32 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 36: number analyzed (Participants) | 1 | 6 | 4 | 1 | 1
  Renal Epithelial Casts Week 36 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.167 (0.4082) | 0.000 (0.0000) | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (NA) — Value was not evaluable because only one participant was analyzed.
  Renal Epithelial Casts Week 40: number analyzed (Participants) | 0 | 4 | 4 | 4 | 2
  Renal Epithelial Casts Week 40 |  | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 44: number analyzed (Participants) | 1 | 5 | 5 | 4 | 2
  Renal Epithelial Casts Week 44 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Renal Epithelial Casts Week 48: number analyzed (Participants) | 2 | 6 | 4 | 3 | 4
  Renal Epithelial Casts Week 48 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Squamous Epithelial Cells Week 1: number analyzed (Participants) | 1 | 4 | 3 | 5 | 3
  Squamous Epithelial Cells Week 1 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.250 (1.2583) | 3.000 (5.1962) | -0.200 (0.4472) | -0.333 (0.5774)
  Squamous Epithelial Cells Week 2: number analyzed (Participants) | 1 | 4 | 4 | 4 | 3
  Squamous Epithelial Cells Week 2 | 1.000 (NA) — Value was not evaluable because only one participant was analyzed. | -8.000 (14.6969) | -0.250 (3.6856) | 0.000 (0.0000) | -1.667 (1.5275)
  Squamous Epithelial Cells Week 4: number analyzed (Participants) | 1 | 3 | 5 | 4 | 2
  Squamous Epithelial Cells Week 4 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | -1.800 (7.1554) | 0.000 (0.0000) | 1.000 (1.4142)
  Squamous Epithelial Cells Week 8: number analyzed (Participants) | 0 | 2 | 4 | 2 | 3
  Squamous Epithelial Cells Week 8 |  | 0.000 (0.0000) | 0.500 (1.0000) | 0.000 (0.0000) | 0.333 (0.5774)
  Squamous Epithelial Cells Week 12: number analyzed (Participants) | 1 | 3 | 5 | 2 | 3
  Squamous Epithelial Cells Week 12 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | -4.333 (7.5056) | -2.200 (5.4955) | 0.000 (0.0000) | 0.333 (0.5774)
  Squamous Epithelial Cells Week 16: number analyzed (Participants) | 1 | 5 | 4 | 5 | 2
  Squamous Epithelial Cells Week 16 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | -2.750 (5.5000) | -0.200 (0.4472) | 0.000 (0.0000)
  Squamous Epithelial Cells Week 20: number analyzed (Participants) | 2 | 4 | 5 | 6 | 4
  Squamous Epithelial Cells Week 20 | 1.000 (1.4142) | -2.750 (5.5000) | -1.400 (5.6391) | -0.167 (0.9832) | -0.750 (0.9574)
  Squamous Epithelial Cells Week 24: number analyzed (Participants) | 0 | 4 | 4 | 7 | 3
  Squamous Epithelial Cells Week 24 |  | 1.000 (1.4142) | 1.000 (2.0000) | -0.286 (0.4880) | 1.333 (4.1633)
  Squamous Epithelial Cells Week 28: number analyzed (Participants) | 1 | 4 | 5 | 4 | 3
  Squamous Epithelial Cells Week 28 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | -3.000 (6.0000) | 0.600 (1.3416) | -0.250 (0.5000) | -1.667 (1.5275)
  Squamous Epithelial Cells Week 32: number analyzed (Participants) | 2 | 2 | 4 | 6 | 2
  Squamous Epithelial Cells Week 32 | 0.500 (0.7071) | 0.000 (0.0000) | 0.500 (1.0000) | -0.667 (0.8165) | -0.500 (0.7071)
  Squamous Epithelial Cells Week 36: number analyzed (Participants) | 1 | 5 | 4 | 1 | 1
  Squamous Epithelial Cells Week 36 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (NA) — Value was not evaluable because only one participant was analyzed.
  Squamous Epithelial Cells Week 40: number analyzed (Participants) | 0 | 4 | 4 | 4 | 2
  Squamous Epithelial Cells Week 40 |  | -2.750 (5.5000) | 0.750 (1.5000) | 0.000 (0.0000) | -0.500 (0.7071)
  Squamous Epithelial Cells Week 44: number analyzed (Participants) | 1 | 5 | 5 | 4 | 2
  Squamous Epithelial Cells Week 44 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | -1.000 (2.2361) | 0.600 (1.3416) | -0.250 (0.5000) | -0.500 (0.7071)
  Squamous Epithelial Cells Week 48: number analyzed (Participants) | 2 | 6 | 4 | 3 | 3
  Squamous Epithelial Cells Week 48 | 0.000 (0.0000) | 0.667 (1.6330) | 1.250 (1.8930) | 0.333 (0.5774) | -1.000 (1.0000)
  Transitional Epithelial Cells Week 1: number analyzed (Participants) | 1 | 4 | 3 | 5 | 3
  Transitional Epithelial Cells Week 1 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 2: number analyzed (Participants) | 1 | 4 | 4 | 4 | 3
  Transitional Epithelial Cells Week 2 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 4: number analyzed (Participants) | 1 | 3 | 5 | 4 | 2
  Transitional Epithelial Cells Week 4 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 8: number analyzed (Participants) | 0 | 3 | 4 | 2 | 3
  Transitional Epithelial Cells Week 8 |  | 1.000 (1.7321) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 12: number analyzed (Participants) | 1 | 3 | 5 | 2 | 3
  Transitional Epithelial Cells Week 12 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.200 (0.4472) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 16: number analyzed (Participants) | 1 | 5 | 4 | 5 | 2
  Transitional Epithelial Cells Week 16 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.400 (0.8944) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 20: number analyzed (Participants) | 2 | 4 | 5 | 6 | 4
  Transitional Epithelial Cells Week 20 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 24: number analyzed (Participants) | 0 | 4 | 4 | 7 | 3
  Transitional Epithelial Cells Week 24 |  | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 28: number analyzed (Participants) | 1 | 4 | 5 | 4 | 3
  Transitional Epithelial Cells Week 28 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 32: number analyzed (Participants) | 2 | 3 | 4 | 6 | 3
  Transitional Epithelial Cells Week 32 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 36: number analyzed (Participants) | 1 | 6 | 4 | 1 | 1
  Transitional Epithelial Cells Week 36 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.167 (0.4082) | 0.000 (0.0000) | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (NA) — Value was not evaluable because only one participant was analyzed.
  Transitional Epithelial Cells Week 40: number analyzed (Participants) | 0 | 4 | 4 | 4 | 2
  Transitional Epithelial Cells Week 40 |  | 0.250 (0.5000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 44: number analyzed (Participants) | 1 | 5 | 5 | 4 | 2
  Transitional Epithelial Cells Week 44 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Transitional Epithelial Cells Week 48: number analyzed (Participants) | 2 | 6 | 4 | 3 | 4
  Transitional Epithelial Cells Week 48 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)

26. Secondary Outcome: Changes From Baseline in Urinalysis Parameters During the Study (Hyaline Casts)
Description: Hyaline casts was measured in cells per low power field (cells/LPF).
Time Frame: as for outcome 13
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: cells/LPF
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 2 | 6 | 5 | 7 | 4
cells/LPF
  Week 1: number analyzed (Participants) | 1 | 4 | 3 | 5 | 3
  Week 1 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 1.000 (1.7321) | -0.200 (0.4472) | 0.000 (0.0000)
  Week 2: number analyzed (Participants) | 1 | 4 | 4 | 4 | 3
  Week 2 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.250 (0.5000) | 1.000 (1.1547) | -0.250 (0.5000) | 0.333 (0.5774)
  Week 4: number analyzed (Participants) | 1 | 3 | 5 | 4 | 2
  Week 4 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | -0.800 (1.0954) | -0.250 (0.5000) | 0.000 (0.0000)
  Week 8: number analyzed (Participants) | 0 | 3 | 4 | 2 | 3
  Week 8 |  | 0.333 (0.5774) | 0.250 (0.5000) | 0.000 (0.0000) | 0.000 (0.0000)
  Week 12: number analyzed (Participants) | 1 | 3 | 5 | 2 | 3
  Week 12 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 5.000 (11.1803) | 0.000 (0.0000) | 0.000 (0.0000)
  Week 16: number analyzed (Participants) | 1 | 5 | 4 | 5 | 2
  Week 16 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.500 (1.0000) | 0.000 (0.0000) | 0.500 (0.7071)
  Week 20: number analyzed (Participants) | 2 | 4 | 5 | 6 | 4
  Week 20 | 0.000 (0.0000) | 0.000 (0.0000) | -0.600 (0.8944) | 1.500 (3.6742) | -0.750 (1.5000)
  Week 24: number analyzed (Participants) | 0 | 4 | 4 | 7 | 3
  Week 24 |  | 0.000 (0.0000) | -0.250 (0.5000) | 0.857 (2.2678) | 0.333 (0.5774)
  Week 28: number analyzed (Participants) | 1 | 4 | 5 | 4 | 3
  Week 28 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | -0.400 (0.8944) | 0.000 (0.0000) | 0.000 (0.0000)
  Week 32: number analyzed (Participants) | 2 | 3 | 4 | 6 | 3
  Week 32 | 0.000 (0.0000) | 0.000 (0.0000) | 1.250 (2.5000) | 0.000 (0.0000) | 13.333 (23.0940)
  Week 36: number analyzed (Participants) | 1 | 6 | 4 | 1 | 1
  Week 36 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.000 (NA) — Value was not evaluable because only one participant was analyzed.
  Week 40: number analyzed (Participants) | 0 | 4 | 4 | 4 | 2
  Week 40 |  | 0.000 (0.0000) | -0.500 (1.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Week 44: number analyzed (Participants) | 1 | 5 | 5 | 4 | 2
  Week 44 | 0.000 (NA) — Value was not evaluable because only one participant was analyzed. | 0.400 (0.8944) | -0.400 (0.8944) | 0.000 (0.0000) | 0.000 (0.0000)
  Week 48: number analyzed (Participants) | 2 | 6 | 4 | 3 | 4
  Week 48 | 0.000 (0.0000) | 1.167 (2.8577) | 0.000 (0.0000) | 0.000 (0.0000) | -0.250 (0.5000)

27. Secondary Outcome: Changes From Baseline in Urinalysis Parameters During the Study (pH)
Description: Urine pH was measured on a pH scale.
Time Frame: as for outcome 13
Population: The SS consisted of all randomized study participants who received at least 1 dose of IMP.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo (SS) | BKZ 16 mg (SS) | BKZ 160 mg (SS) | BKZ 160 mg LD (SS) | BKZ 320 mg (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 41 | 41
pH
  Week 1: number analyzed (Participants) | 40 | 38 | 43 | 41 | 40
  Week 1 | -0.138 (0.9198) | 0.197 (0.5875) | 0.023 (0.8014) | 0.085 (0.6011) | 0.000 (0.8321)
  Week 2 | -0.155 (0.9072) | 0.154 (0.7708) | -0.081 (0.7149) | 0.134 (0.8293) | -0.012 (0.7541)
  Week 4: number analyzed (Participants) | 41 | 38 | 41 | 40 | 41
  Week 4 | -0.195 (0.9211) | 0.026 (0.6571) | -0.134 (0.8368) | 0.063 (0.6620) | -0.098 (0.6729)
  Week 8: number analyzed (Participants) | 41 | 39 | 42 | 38 | 41
  Week 8 | 0.000 (0.7826) | 0.077 (0.7393) | -0.024 (0.8762) | 0.263 (0.7235) | 0.024 (0.7579)
  Week 12: number analyzed (Participants) | 40 | 38 | 43 | 38 | 41
  Week 12 | -0.100 (1.0203) | 0.237 (0.7600) | -0.047 (0.6971) | 0.211 (0.6641) | 0.073 (0.8843)
  Week 16: number analyzed (Participants) | 42 | 38 | 41 | 38 | 40
  Week 16 | -0.107 (0.8449) | 0.092 (0.7957) | -0.122 (0.8199) | 0.118 (0.7207) | 0.088 (0.7240)
  Week 20: number analyzed (Participants) | 40 | 39 | 42 | 37 | 40
  Week 20 | -0.113 (0.7884) | 0.269 (0.8649) | -0.012 (0.8300) | -0.054 (0.6539) | 0.063 (0.8929)
  Week 24: number analyzed (Participants) | 39 | 38 | 41 | 35 | 39
  Week 24 | -0.154 (0.9400) | -0.013 (0.8011) | -0.085 (0.6605) | 0.100 (0.4820) | -0.026 (0.6973)
  Week 28: number analyzed (Participants) | 39 | 38 | 41 | 35 | 40
  Week 28 | -0.090 (0.8419) | -0.053 (0.6657) | -0.122 (0.7313) | 0.086 (0.6122) | -0.088 (0.6783)
  Week 32: number analyzed (Participants) | 39 | 38 | 40 | 34 | 39
  Week 32 | -0.218 (0.8335) | -0.079 (0.7491) | 0.063 (0.8784) | -0.103 (0.6717) | -0.269 (0.5718)
  Week 36: number analyzed (Participants) | 38 | 38 | 41 | 34 | 39
  Week 36 | -0.211 (0.8353) | 0.118 (0.7300) | -0.195 (0.8506) | -0.118 (0.6038) | -0.077 (0.7569)
  Week 40: number analyzed (Participants) | 37 | 37 | 40 | 34 | 39
  Week 40 | -0.216 (0.9394) | -0.041 (0.6388) | -0.188 (0.8525) | -0.191 (0.5643) | -0.154 (0.7448)
  Week 44: number analyzed (Participants) | 36 | 38 | 41 | 33 | 38
  Week 44 | -0.458 (0.7780) | -0.171 (0.7002) | -0.159 (0.9044) | -0.167 (0.6693) | -0.171 (0.7285)
  Week 48: number analyzed (Participants) | 38 | 36 | 40 | 33 | 40
  Week 48 | -0.092 (1.0771) | -0.014 (0.7318) | -0.200 (0.8533) | -0.015 (0.7855) | -0.100 (0.7528)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Baseline until the Safety Follow-Up Visit (up to Week 68)
Description: At Week 12, Placebo and BKZ 16 mg subjects were re-randomized to either BKZ 160 mg or BKZ 320 mg. Subjects randomized to BKZ 160 mg or BKZ 320 mg at Baseline were not re-randomized at Week 12 and remained on their treatment. The Safety Set is based on actual treatment, other populations are based on planned treatment. 160mg LD is considered 160mg.
Arm/Group | Placebo (SS) - up to Wk 12 | BKZ 16 mg (SS) - up to Wk 12 | BKZ 160 mg & 160 mg LD (SS) - up to Wk 68 | BKZ 320 mg (SS) - up to Wk 68
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39 | 0/126 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/39 | 8/126 | 0/80
Other Adverse Events (participants affected / at risk) | 8/42 | 9/39 | 40/126 | 29/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) - up to Wk 12 (N=42) | BKZ 16 mg (SS) - up to Wk 12 (N=39) | BKZ 160 mg & 160 mg LD (SS) - up to Wk 68 (N=126) | BKZ 320 mg (SS) - up to Wk 68 (N=80)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) - up to Wk 12 (N=42) | BKZ 16 mg (SS) - up to Wk 12 (N=39) | BKZ 160 mg & 160 mg LD (SS) - up to Wk 68 (N=126) | BKZ 320 mg (SS) - up to Wk 68 (N=80)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 8 (8) | 2 (3)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 7 (8) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 12 (15) | 11 (11)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 12 (12) | 8 (10)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Biomarker assays were not rigorously validated, thus it was not possible to use results for PD as a secondary objective. The results were interpreted with caution for exploratory purpose, and thus are not shared in this report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT02969525/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT02969525/SAP_001.pdf